# Evaluation of the Safety, Tolerability, Efficacy and Activity of AMX0035, a Fixed Combination of Phenylbutyrate (PB) and Tauroursodeoxycholic Acid (TUDCA), for Treatment of Amyotrophic Lateral Sclerosis (ALS)

**Regulatory Sponsor:** Amylyx Pharmaceuticals Inc.

**Funding Sponsor:** Amylyx Pharmaceuticals Inc.

**Study Product:** AMX0035

**Protocol Number:** AMX3500

**IND Number:** 129563

**Draft or Version Number:** 7.0

30 Mar 2020

The information contained herein is confidential and proprietary in nature, and will not be disclosed to any third party without written approval of authorized designee.

This document may be disclosed to the appropriate institutional review boards or to duly authorized representatives of the US Food and Drug Administration or a national regulatory authority under the condition that they maintain confidentiality.

AMX-0035 in ALS

Protocol Number: AMX3500

Version 7.0

#### STATEMENT OF COMPLIANCE

This study will be conducted in compliance with the protocol, International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH), Good Clinical Practice (GCP), and the applicable regulatory requirements, United States Code of Federal Regulations (CFR) Title 45 CFR Part 46 and Title 21 CFR Parts 50, 56, and 312.

AMX-0035 in ALS Protocol Number: AMX3500 Version 7.0

#### SIGNATURE PAGE

I have read the attached protocol entitled, Evaluation of the Safety, Tolerability, Efficacy and Activity of AMX0035, a Fixed Combination of Phenylbutyrate (PB) and Tauroursodeoxycholic Acid (TUDCA), for Treatment of Amyotrophic Lateral Sclerosis (ALS) dated March 30, 2020 (Version 7.0) and agree to abide by all described protocol procedures. I agree to comply with the International Conference on Harmonisation Tripartite Guideline on Good Clinical Practice, applicable FDA regulations and guidelines identified in 21 CFR Parts 11, 50, 54, and 312, Institutional Review Board (IRB) and local institutional guidelines and policies, and the Health Insurance Portability and Accountability Act (HIPAA).

| Site Investigator: | |
|--------------------|-------|
| Signed: | Date: |


## TABLE OF CONTENTS

| ST | <b>TATE</b> | EMENT OF COMPLIANCE ····· | 2 |
|---|---|---|---|
| SI | GNA | ATURE PAGE ···· | 3 |
| LI | ST C | OF ABBREVIATIONS | 8 |
| ΡI | ROTO | OCOL SUMMARY ······ | 10 |
| | | DULE OF ACTIVITIES | |
| | | Y WORKFLOW ······ | |
| <b>S</b> 1 | | | |
| 1 | E | THICS/PROTECTION OF HUMAN SUBJECTS ····· | |
| | 1.1 | INSTITUTIONAL REVIEW BOARD (IRB) · | 16 |
| | 1.2 | ETHICAL CONDUCT OF STUDY | |
| | 1.3 | SUBJECT INFORMATION AND CONSENT | 16 |
| 2 | II | NTRODUCTION: BACKGROUND INFORMATION AND SCIENTIFIC RATIONALE······ | 17 |
| | 2.1 | BACKGROUND INFORMATION | 17 |
| | | 2.1.1 ALS Overview | |
| | | 2.1.2 AMX0035 Rationale ····· | |
| | | 2.1.3 Prior Clinical Use of PB and TUDCA in Subjects with ALS····· | 18 |
| | | 2.1.4 Additional Previous Clinical Experience with Phenylbutyrate · | 21 |
| | | 2.1.5 Additional Previous Clinical Experience with TUDCA | 25 |
| | | 2.1.6 Previous Clinical Experience with Ursodiol (UDCA)····· | 30 |
| | 2.2 | POTENTIAL RISKS AND BENEFITS | |
| | | 2.2.1 Potential Risks | |
| | | 2.2.2 Known Potential Benefits | |
| 3 | O | OBJECTIVES ····· | |
| | 3.1 | STUDY OBJECTIVES ···· | |
| | 3.2 | STUDY OUTCOME MEASURES ····· | |
| | | 3.2.1 Primary Outcome Measures ····· | 34 |
| | | 3.2.2 Secondary Outcome Measures ····· | 35 |
| 4 | S | TUDY DESIGN | 36 |
| | 4.1 | OVERALL STUDY DESIGN AND PLAN····· | |
| | 4.2 | STUDY CENTERS | 36 |
| | 4.3 | STUDY DURATION | |
| | 4.4 | PROTOCOL ADHERENCE ···· | 36 |
| 5 | S | TUDY ENROLLMENT AND WITHDRAWAL······ | 37 |
| | 5.1 | NUMBER OF STUDY SUBJECTS ···· | |
| | 5.2 | INCLUSION AND EXCLUSION CRITERIA | |
| | | 5.2.1 Inclusion Criteria | |
| | | 5.2.2 Exclusion Criteria | |
| | 5.3 | TREATMENT ASSIGNMENT PROCEDURES · | 41 |

AMX-0035 in ALS

Protocol Number: AMX3500


| | 5.3.1 Randomization Procedures · | |
|---|---|---|
| 5.4 | | |
| | 5.4.1 Handling of Withdrawals | |
| 5.5 | TERMINATION OF STUDY · | 43 |
| 6 | TREATMENTS ADMINISTERED ····· | ····· <b>4</b> 4 |
| <b>6</b> .1 | | |
| | 6.1.1 Study Product Description | |
| | 6.1.2 Placebo Placebo | |
| 6.2 | | |
| | 6.2.1 Formulation, Packaging, and Labeling ····· | 46 |
| | 6.2.2 Product Storage and Stability | 46 |
| | 6.2.3 Dispensing Product | |
| 6.3 | 47 | |
| | 6.3.1 Feeding Tube Study Drug Administration | 48 |
| 6.4 | MODIFICATION OF STUDY INTERVENTION/INVESTIGATIONAL PRODUCT FOR A SUBJECT ······· | 48 |
| | 6.4.1. Dosage Discontinuation | 48 |
| 6.5 | | 49 |
| 6.6 | | |
| <b>6.7</b> | | |
| | 6.7.1 Prohibited Medications and Contraindications ····· | 50 |
| 7 : | STUDY SCHEDULE····· | 52 |
| 7.1 | | |
| 7.2 | | |
| | 7.2.1 Screen Failures | |
| 7.3 | | 53 |
| 7.4 | BASELINE VISIT · | 54 |
| 7.5 | | |
| 7.6 | | |
| 7.7 | WEEK 9 TELEPHONE VISIT ····· | 55 |
| 7.8 | WEEK 12 CLINIC VISIT····· | 56 |
| 7.9 | WEEK 15 PHONE VISIT ····· | 56 |
| 7.1 | 0 Week 18 Clinic Visit · | 57 |
| 7.1 | | 57 |
| 7.13 | | 57 |
| 7.13 | | 58 |
| 7.1 | | |
| 7.1 | | |
| 7.1 | 6 PROTOCOL DEVIATIONS | 59 |
| | 7.16.1 Missed Visits and Procedures ····· | 59 |
| 7.1 | | |
| 0 | CLINICAL ACCECCMENTS AND OUTCOME MEASURES | |
| 8 | CLINICAL ASSESSMENTS AND OUTCOME MEASURES | 61 |
| 81 | CLINICAL VARIARIES | 61 |

Protocol Number: AMX3500


| | 8.1.1 | Vital Signs, Height & Weight ····· | 61 |
|---|---|---|---|
| | 8.1.2 | Clinical Laboratory Assessments · | 61 |
| | 8.1.3 | Biomarkers and Pharmacokinetic Analysis ····· | 62 |
| | 8.1.4 | Blood Samples for Future Research Use | |
| | | 2-Lead Electrocardiogram (ECG) · | 63 |
| | 8.1.6 | Physical Examination | |
| | 8.1.7 | Neurological Examination | |
| | 8.1.8 | Upper Motor Neuron-Burden (UMN-B) | 63 |
| | 8.1.9 | Columbia Suicide Severity Rating Scale (C-SSRS) | 63 |
| | 8.1.10 | Exit Questionnaire | |
| | | Adverse Events····· | |
| 8.2 | OUTCO | DME MEASURES · | |
| | 8.2.1 | ALSFRS-R (Amyotrophic Lateral Sclerosis Functional Rating Scale – Revised)······ | 64 |
| | 8 <b>.2.2</b> | Pulmonary Function Testing - Slow Vital Capacity (SVC) | 64 |
| | 8.2.3 | Isometric Strength Testing (ATLIS) ····· | 65 |
| | 8.2.4 | Neuroimaging MR-PET Sub-Study ····· | |
| | 8.2.5 Su | ırvival Assessment | |
| | 8.2.6 | Training and Validation ····· | 65 |
| 0 0 | A DECES | AND ADVERSE EVENTS ····· | (1 |
| 9 S | AFEIY | AND ADVERSE EVENTS | 00 |
| 9.1 | DEFINI | TIONS OF AES, SUSPECTED ADVERSE DRUG REACTIONS & SAES ····· | 66 |
| | 9.1.1 | Adverse Event and Suspected Adverse Drug Reactions | 66 |
| | 9.1.2 | Serious Adverse Events | 67 |
| 9.2 | | SMENT AND RECORDING OF ADVERSE EVENTS | |
| > <b></b> | 9.2.1 | Assessment of Adverse Events | 65 |
| | 9.2.2 | Relatedness of Adverse Event to Investigational Product | |
| | | dverse Events in Prior Human Experience with Each Individual Component | 70 |
| | 9.2.4 | Recording of Adverse Events | 70 |
| 9.3 | | SE EVENTS AND SERIOUS ADVERSE EVENTS - REPORTABLE EVENTS | 7( |
| 10 D | ATA A | ND SAFETY MONITORING AND STATISTICAL ANALYSIS PLAN ······ | 72 |
| 10.1 | Вля | TA AND SAFETY MONITORING BOARD | |
| | | TISTICAL CONSIDERATIONS | |
| 10.2 | | | |
| | 10.2.1 | Statistical Methods | |
| | 10.2.2 | Analysis for Safety Analysis for Efficacy | ····· 73 |
| | 10.2.3 | Analysis for Efficacy Analysis Populations | |
| 40.0 | 10.2.4 | | |
| 10.3 | MIS | SING DATA | 72 |
| 11 D | ATA CO | OLLECTION, MANAGEMENT AND MONITORING | 75 |
| 11.1 | Roi | LE OF DATA MANAGEMENT · | |
| | 11.1.1 | Data Entry and Checks | |
| | 11.1.2 | Data Lock Process ···· | |
| | 11.1.3 | Quality Assurance | |
| 11.2 | CLI | NICAL MONITORING | ····· 76 |
| 11.3 | DAT | A HANDLING AND RECORD KEEPING ····· | ····· 76 |
| | 11.3.1 | Confidentiality | |
| | 11.3.2 | Study Discontinuation | 76 |
| | | v | |

Protocol Number: AMX3500


| | 11.3.3 | Retention of Records | 77 |
|---|---|---|---|
| | 11.3.4 | Publications | 77 |
| 12 | LITERAT | TURE REFERENCES····· | <b>78</b> |
| 13 | APPEND | ICES { | <b>30</b> |
| | 13.1 APPEND | IX I: EL ESCORIAL WORLD FEDERATION OF NEUROLOGY CRITERIA FOR THE DIAGNOSIS OF ALS $\cdots$ { | 30 |
| | 13.2 APPENI | DIX II: ALS FUNCTIONAL RATING SCALE – REVISED (ALSFRS-R) · | 32 |
| | 13.3 APPENI | DIX III: COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS) BASELINE VERSION · | 35 |
| | 13.4 APPENI | DIX IV: COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS) SINCE LAST VISIT VERSION · | 38 |
| | 13.5 APPENI | DIX V: CENTER FOR NEUROLOGICAL STUDY – LABILITY SCALE ······ | 91 |
| | | DIX VI: INSTRUCTIONS TO PATIENTS | |
| | 13.7 APPEN | IDIX VII: AMX-0035 IN ALS OPEN LABEL EXTENSION (OLE): | 93 |

AMX-0035 in ALS Protocol Number: AMX3500 Version 7.0 Version date 30Mar2020

#### LIST OF ABBREVIATIONS

ADR Adverse Drug Reaction

AE Adverse Event/Adverse Experience

b.i.d Twice a Day

CFR Code of Federal Regulations
CIB Clinical Investigator's Brochure
cIRB Central Institutional Review Board

CRF Case Report Form

DSMB Data and Safety Monitoring Board eCRF Electronic Case Report Form ER Endoplasmic Reticulum FDA Food and Drug Administration

EWA Endand wide Assumence

FWA Federal-wide Assurance

g Gram

GCP Good Clinical Practice
GUID Globally Unique Identifier

HIPAA Health Insurance Portability and Accountability Act

ICF Informed Consent Form

ICH International Conference on Harmonisation

IDE Investigational Device Exemption
IND Investigational New Drug Application

IRB Institutional Review Board ITT Modified Intent to Treat MOP Manual of Procedures

MPRAGE Magnetization Prepared Rapid Gradient Echo

N Number (typically refers to subjects)

NDA New Drug Application NYGC New York Genome Center NIH National Institutes of Health

OHRP Office for Human Research Protections
OHSR Office of Human Subjects Research

OLE Open Label Extension

PAA Phenylacetate (metabolite of PB)

PB Sodium Phenylbutyrate

PET Positron Emission Tomography

PCP Primary Care Provider

PHI Protected Health Information

PI Principal Investigator
QA Quality Assurance
QC Quality Control

AMX-0035 in ALS

Protocol Number: AMX3500


ROI Region of Interest

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan

SI Site Investigator

SMC Safety Monitoring Committee SOP Standard Operating Procedure

SUSAR Suspected Unexpected Serious Adverse Reaction

t.i.d Three Times a Day

UDCA Ursodeoxycholic Acid (ursodiol)
TUDCA Tauroursodeoxycholic Acid

US United States

AMX-0035 in ALS

Protocol Number: AMX3500


#### PROTOCOL SUMMARY

#### **Study Title**

Evaluation of the Safety, Tolerability, Efficacy and Activity of AMX0035, a Fixed Combination of Phenylbutyrate (PB) and Tauroursodeoxycholic Acid (TUDCA), for Treatment of Amyotrophic Lateral Sclerosis (ALS)

## Version Number

4.0

#### **Study Indication**

Amyotrophic Lateral Sclerosis (ALS)

#### **Phase of Development**

II

#### **Rationale for the Study**

The objective of this study is to determine the safety and efficacy of AMX0035 in subjects with Amyotrophic Lateral Sclerosis (ALS). ALS is a progressive neurodegenerative disease for which there is no cure. There are only two medications approved specifically for treating ALS. This includes Rilutek (riluzole), which only provides a modest benefit for subjects, and Radicava (edaravone). ALS also exacts a significant economic burden.

AMX0035 has demonstrated efficacy in models of neurodegeneration, classical activation of neuroinflammation, and bioenergetics deficits. The individual components of AMX0035, PB and TUDCA have demonstrated efficacy in *in vivo* models of ALS, Parkinson's, Alzheimer's, ischemia, and many others. Each individual component has also been tested in small clinical trials of ALS subjects and was found to be safe and well-tolerated, and hit primary endpoints of efficacy.

The first trial under this IND will be a randomized double-blind placebo-controlled Phase II trial to evaluate the safety and efficacy of AMX0035 for treatment of ALS. The program is designed to demonstrate that treatment is safe, can slow the decline in function, muscle strength, and vital capacity, and to assess the impact of AMX0035 therapy on biomarkers of ALS including blood levels of phosphorylated axonal neurofilament H subunit and 18 kDa translocator protein PET tracer uptake. This Phase II trial would also serve as the basis for the design of a pivotal trial in this subject population.

#### **Study Design**

This is a multicenter, randomized, double-blind, placebo-controlled 28-week study evaluating the safety, tolerability, efficacy, pharmacokinetics and biological activity of AMX0035.

AMX-0035 in ALS

Protocol Number: AMX3500


#### **Study Objectives and Endpoints**

The primary objective of the study is to assess safety, tolerability, and efficacy of oral (or feeding tube) administration of AMX0035 via sachet (3g PB and 1g TUDCA) twice daily vs. matched placebo administered via sachet twice daily.

The primary outcome measures will be:

- 1. To confirm the safety and tolerability of AMX0035 in subjects with ALS over a 24-week period
- 2. To measure the impact of treatment on disease progression using the slope of the revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R)

The secondary objectives of the study will be:

- 1. To assess the impact of AMX0035 on the rate of decline of isometric muscle strength, as measured by the Accurate Test of Limb Isometric Strength (ATLIS)
- 2. To assess the impact of AMX0035 on disease progression as measured by Slow Vital Capacity (SVC) decline, time to tracheostomy, and survival
- 3. To assess the impact of AMX0035 on biomarkers including blood levels of phosphorylated axonal neurofilament H subunit (pNF-H) and 18 kDa translocator protein (TSPO) PET tracer uptake
- 4. To determine the population pharmacokinetics parameters of PB and TUDCA at steady state during treatment with AMX0035
- 5. To measure the impact of the treatment on survival.

#### **Study Locations**

Up to 25 Northeast ALS Consortium (NEALS) centers in the United States will participate in the study.

#### **Number of Planned Subjects**

Approximately 132 subjects will be randomized in the study.

#### **Study Population**

This study will be conducted in subjects who have sporadic or familial ALS diagnosed as definite as defined by revised El Escorial criteria (Appendix 1). Subjects must provide written informed consent prior to screening. At screening, eligible subjects must be at least 18 years old and less than 80 years old, and have a  $VC \ge 60\%$  of predicted capacity for age, height and gender. Subjects must have had onset of ALS symptoms less than or equal to 18 months prior to the screening visit, defined as first onset of weakness. Subjects on a stable dose of riluzole and those not taking riluzole, and women of child-bearing age at screening are eligible for inclusion as long as they meet specific protocol requirements. There will be no restrictions for subjects taking Radicava (edaravone) at the time of screening, or if started while enrolled in the study. Detailed criteria are described in the body of the protocol.

AMX-0035 in ALS

Protocol Number: AMX3500


## **Treatment Groups**

Subjects will be randomly assigned in a 2:1 ratio to oral (or feeding tube) AMX0035 treatment (1 sachet= 3g PB and 1g TUDCA plus excipients) or matching placebo. For the first three weeks of dosing, subjects will take one sachet daily (i.e. half-dose) and if tolerated will increase to two sachets daily.

## **Duration of Treatment and Follow-up**

Subjects will remain on treatment until the Week 24 visit. Each randomized subject will also have a Final Telephone Interview 28 days (+ 5 days) after last dose of study drug to assess for adverse events (AEs), changes in concomitant medications and to administer the ALSFRS-R.

# SCHEDULE OF ACTIVITIES

| | | | | | Study | Drug Adm | inistration ( | (weeks) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ACTIVITY | Screening<br>Visit | Baseline<br>Visit <sup>1</sup> | Week 3 | Week 6 | Week 9 | Week<br>12 | Week<br>15 | Week<br>18 | Week 21 | Week 24 OR<br>Early<br>Discontinuation/<br>Final Safety Visit | Final Follow-<br>up Telephone<br>Call <sup>2</sup> | MR-PET Sub-<br>Study Subjects<br>Only |
| | Clinic | Clinic | Clinic | Clinic | Phone | Clinic | Phone | Clinic | Phone | Clinic | Phone | At MGH |
| | -42 Days | Day 0 | Day 21<br>±5 | Day 42<br>±5 | Day 63<br>±5 | Day 84<br>±5 | Day 105<br>±5 | Day<br>126 ±5 | Day 147<br>±5 | Day 168 ±5 | 28 +5 days | |
| Written Informed Consent | X | | | | | | | | | | | X |
| Inclusion/Exclusion Review | X | X | | | | | | | | | | X |
| Medical History<br>History/Demographics | X | | | | | | | | | | | |
| ALS Diagnosis/ALS History | X | | | | | | | | | | | |
| Vital Signs <sup>3</sup> | X | X | X | X | | X | | X | | X | | |
| Neurological Exam <sup>4</sup> | X | | | | | X | | | | X | | $X^4$ |
| Physical Exam <sup>5</sup> | X | | | | | X | | | | X | | |
| Blood Draw for Safety Labs <sup>6</sup> | X | X | X | X | | X | | X | | X | | |
| Blood Draw for Serum Pregnancy<br>Test for WOCB <sup>6</sup> | X | | | | | | | | | | | |
| Urine Sample for Urinalysis <sup>6</sup> | X | X | X | X | | X | | X | | X | | |
| 12-Lead ECG | X | | | | | X | | | | X | | |
| ALSFRS-R | X | X | X | X | X | X | X | X | X | X | X | X |
| Slow Vital Capacity | X | X | | X | | X | | X | | X | | |
| ATLIS Testing | X | X | | X | | X | | X | | X | | |
| Columbia-Suicide Severity Scale <sup>7</sup> | | $X^7$ | X | X | | X | | X | | X | | |
| Exit Questionnaire | | | | | | | | | | X | | |
| MR-PET Scan <sup>8</sup> | | X | | | | | | X | | | | X <sup>8</sup> |
| Blood draw for Biomarker Testing <sup>9</sup> | | X | | X | | X | | X | | X | | |
| Blood draw for PK Analysis <sup>10</sup> | | X | | | | X | | | | X <sup>11</sup> | | |
| Blood draw for optional DNA collection <sup>12</sup> | | X | X | X | | X | | X | | X | | |
| Adverse Events <sup>13</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| Blood draw for TSPO affinity testing <sup>14</sup> | X | | | | | | | | | | | |
| Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X | X |
| Randomization <sup>15</sup> | | X | | | | | | | | | | |
| Dispense Study Drug <sup>16</sup> | | X | | X | | X | | X | | | | |
| Drug Accountability/ Compliance | | | $X^{17}$ | X | X | X | X | X | X | X | | |

AMX-0035 in ALS

Protocol Number: AMX3500


<sup>&</sup>lt;sup>1</sup>The Baseline Visit should occur no more than 42 days after the Screening Visit.

<sup>&</sup>lt;sup>2</sup>A Final Safety Telephone Call will be conducted 28 (+5 days) after the subject takes their last dose of study drug (whether or not the subject has discontinued from the study) to assess for adverse events (AEs), changes in concomitant medications and to administer the ALSFRS-R. This call will only be required for subjects who do NOT enroll in the OLE.

<sup>&</sup>lt;sup>3</sup>Vital signs include systolic and diastolic pressure in mmHg, respiratory rate/minute, heart rate/minute and temperature.

<sup>&</sup>lt;sup>4</sup> The standard Neurological Exam will be used for all patients. The Upper Motor Neuron Burden Scale (UMN-B) will be included for the MR-PET Sub-Study only and administered at the time of the scan.

<sup>&</sup>lt;sup>5</sup>Physical Exam will include height and weight. Height will be collected at Screening Visit ONLY.

<sup>&</sup>lt;sup>6</sup>Safety labs include Hematology (CBC with differential), Complete Chemistry Panel, Liver Function Tests and Urinalysis. Serum pregnancy testing will occur in women of child bearing potential (WOCBP) at the Screening Visit and as necessary during the course of the study.

<sup>&</sup>lt;sup>7</sup>C-SSRS Baseline version to be completed at Baseline Visit only. C-SSRS Since Last Visit version to be completed at all other visits.

<sup>&</sup>lt;sup>8</sup>Approximately 20 subjects will receive MR-PET (Magnetic Resonance-Positron Emission Tomography) scanning completed at selected sites. First scan will occur PRIOR to the Baseline Visit (pre-dose) and the second scan will occur between the Week 12 and Week 21 study visits. MR-PET subjects will also provide blood samples for peripheral blood mononuclear cell (PBMC) extraction prior to each MR-PET scan.

<sup>&</sup>lt;sup>9</sup>Subjects will provide a blood sample for biomarker testing and storage in a biorepository.

<sup>&</sup>lt;sup>10</sup>All subjects will provide a blood sample for pharmacokinetic (PK) testing at the Baseline Visit (pre-dose). Subjects will also provide a blood sample either 1 hour or 4 hours post-dose (±10 minute window per time point) at the Week 12 and Week 24 Visits. PK times will be randomized such that every subject has a 1-hour draw at one visit and a 4-hour draw at the other.

<sup>&</sup>lt;sup>11</sup>PK should not be drawn for early termination subjects

<sup>&</sup>lt;sup>12</sup> If Baseline visit has already occurred or the sample was not collected, DNA should be obtained at next available visit. This is a one-time collection.

<sup>&</sup>lt;sup>13</sup>Adverse events that occur AFTER signing the consent form will be recorded.

<sup>&</sup>lt;sup>14</sup>For MR-PET Sub-Study subjects only, blood will be drawn for TSPO testing at the subject's site during the Screening Visit.

<sup>&</sup>lt;sup>15</sup>Randomization should occur at the Baseline Visit. Randomization will entail entering a subject's kit number into the data capture system.

<sup>&</sup>lt;sup>16</sup>First dose of study drug will be administered in clinic after ALL Baseline Visit procedures are completed.

<sup>&</sup>lt;sup>17</sup>Notify subjects of increase from one sachet per day to two sachets per day

## STUDY WORKFLOW





Subjects who discontinue from the study early will be asked to return to the study site for Final Safety Assessments

AMX-0035 in ALS

Protocol Number: AMX3500


#### 1 ETHICS/PROTECTION OF HUMAN SUBJECTS

## 1.1 Institutional Review Board (IRB)

This study will be conducted in compliance with current Good Clinical Practices (GCP) and Title 21 Part 56 of the United States of America Code of Federal Regulations (CFR) relating to IRBs.

#### 1.2 Ethical Conduct of Study

The study will be conducted in accordance with GCP defined by the International Conference on Harmonization (ICH) and the ethical principles of the Declaration of Helsinki.

## 1.3 Subject Information and Consent

This study will be conducted in compliance with Title 21 Part 50 of the United States of America Code of Federal Regulations (CFR), Federal Regulations and ICH Guidance Documents pertaining to informed consent. At the first visit, prior to initiation of any study-related procedures, subjects will be informed about the nature and purpose of the study, participation/termination conditions, and risks and benefits. Subjects will be given adequate time to ask questions and become familiar with the study prior to providing consent to participate. Subjects will give their written consent to participate in the study and will be provided with a copy of the fully executed consent form for their records.


## 2 Introduction: Background Information and Scientific Rationale

## 2.1 Background Information

#### 2.1.1 ALS Overview

ALS is the most prevalent, adult-onset, progressive motor neuron disease, affecting more than 20,000 subjects in the US and an estimated 450,000 people worldwide, according to the ALS Association. ALS causes the progressive degeneration of motor neurons, resulting in rapidly progressing muscle weakness and atrophy that eventually leads to partial or total paralysis; on average, the disease is fatal within just 3-5 years. There are two FDA-approved medications for ALS, riluzole, which only extends survival modestly, and Radicava (edaravone). ALS also exacts a significant economic burden.

Although the precise cause of ALS is unknown, ALS and other neurodegenerative diseases such as Alzheimer's are strongly characterized by nerve cell death and inflammation. Together these processes form a toxic cycle that is a key driver of progressive neurological decline. Recent research has highlighted mitochondrial stress and endoplasmic reticulum (ER) stress as key mediators of both the nerve cell death and neuroinflammatory processes<sup>1</sup>. The mitochondrion is the energy production center of the cell, while the ER is the quality control center. These two organelles are in constant communication, and are in fact physically connected by a membrane, and their health is vital to cell survival. When either of these cellular processes goes awry, the resulting stress can either kill the cell and/or create inflammation. The brain is extremely sensitive to both mitochondrial stress and ER stress, and both of these pathways have been strongly implicated in causing neurodegenerative disease. We believe that only therapeutically targeting both organelles simultaneously will enact a significant and lasting benefit.

#### 2.1.2 AMX0035 Rationale

AMX0035 is a proprietary combination of two small molecules, phenylbutyrate (PB) and tauroursodeoxycholic acid (TUDCA), designed to block neuronal death and neurotoxic inflammation through simultaneous inhibition of endoplasmic reticulum (ER) stress and mitochondrial stress.

Both PB and TUDCA have been evaluated individually in many disease-specific models of ALS and other neurodegenerative diseases, and in many nonspecific models of ER Stress and bioenergetic stress, respectively.

PB is a pan-HDAC inhibitor and ameliorates ER stress through upregulation of the master chaperone regulator DJ-1 and through recruitment of other chaperone proteins<sup>2</sup>,3. The large increase in chaperone production reduces activation of canonical ER stress pathways, folds misfolded proteins, and has been shown to increase survival in many in vivo models including

AMX-0035 in ALS

Protocol Number: AMX3500


the G93A SOD1 mouse model of ALS<sup>4</sup>. Phenylbutyrate has also been effective in additional in vivo models of Huntington's Disease, Alzheimer's, and Parkinson's <sup>5,6,7</sup>.

TUDCA recovers mitochondrial bioenergetic deficits through incorporating into the mitochondrial membrane, reducing Bax translocation to the mitochondrial membrane, reducing mitochondrial permeability, and increasing the apoptotic threshold of the cell<sup>8</sup>. TUDCA has exhibited efficacy in many in vivo oxidative insult models, including mouse models of stroke, retinal disease, cardiac disease, brain lipopolysaccharide insult, the MPTP mouse model of Parkinson's, and ALS in vitro models of poly(GA)-induced toxicity<sup>9,10,11</sup>.

Either ER stress or bioenergetic stress can result in neuronal death and a cytotoxic immune response. We therefore combined PB and TUDCA and have since demonstrated that they have synergistic efficacy when dosed in particular ratios. The combination of agents demonstrated a mathematically synergistic increase in neuronal viability in a strong oxidative insult model (H2O2-mediated toxicity) by linear modeling.

Cytotoxic neuroinflammation has been found to be a major part of neurodegeneration<sup>12,13,14</sup>. Different ratios of AMX0035 reduced classical activation of cytotoxic cytokines and increased phagocytic cytokines in an LPS-insult, glial model of inflammation.

#### 2.1.3 Prior Clinical Use of PB and TUDCA in Subjects with ALS

Both PB and TUDCA have been evaluated in subjects with ALS and were found to be safe, well-tolerated, and exhibited preliminary signs of efficacy. PB was evaluated in a 20-week safety and biomarker study in ALS subjects<sup>15</sup>. This was a Phase I dose escalation trial and each subject was scheduled to receive PB at increasing dose from 9 to 21 g/day. A total of 40 subjects were recruited at 8 sites in the US. Twenty-six subjects completed the 20-week treatment phase. Histone acetylation was decreased by approximately 50% in blood buffy-coat specimens at screening and was significantly increased after PB administration. Blood levels of PB and the primary metabolite, phenylacetate, increased with dosage (Figure 1) with a plateau between the 3 and 6 gram t.i.d. regimen. While the majority of subjects tolerated higher dosages of PB, the lowest dose (9 g/day), was the most effective at increasing histone acetylation levels in blood (Figure 2). Treatment with PB did not alter blood riluzole levels. Adverse events in subjects taking riluzole and NaPB together did not occur more frequently, compared to those on PB alone.




**Figure 1**: Histone acetylation levels with PB dose. Blood histone acetylation levels are shown compared with dose taken prior to blood draw. The error bars represent standard error. (Doses are repeated t.i.d in this study)



**Figure 2**: Phenylbutyrate and phenylacetate levels. Blood phenylbutyrate and phenylacetate levels are shown compared with dose taken prior to blood draw. The error bars represent standard error (doses are repeated t.i.d in this study).

Protocol Number: AMX3500


It is not clear why acetylation levels were highest at 9 g/day. However, the author noted that in a study of PB in Huntington's disease, the effects of PB on mRNA expression levels of a 12-gene biomarker set were greatest at lowest dosages (4 g t.i.d.) with an inverse dose response<sup>16</sup>.

For the planned Phase II trial of PB in combination with TUDCA, we therefore selected a dose of 3 grams of PB twice a day (6 grams per day) as a target dose with the desired pharmacologic effect.

Recently, TUDCA at 1g b.i.d. demonstrated a statistically significant slowing of ALSFRS-R progression rate in a year-long, multi-site, placebo-controlled clinical trial of ALS<sup>17</sup>. In this proof-of-principle trial, 34 ALS subjects under treatment with riluzole were randomized to placebo or TUDCA (1 gram b.i.d.) for 54 weeks. The proportion of responders (defined as subjects with >15% improvement in ALSFRS-R slope) was higher under TUDCA (87%) than under placebo (P = 0.021; 43%). At study end, baseline-adjusted ALSFRS-R was significantly higher (P = 0.007) in TUDCA than in placebo groups. Comparison of the slopes of regression analysis showed slower progression in the TUDCA than in the placebo group (P < 0.01) (Figure 3).



**Figure 3**: Linear regression analysis of ALSFRS-R mean scores over time for the TUDCA (circles, slope -0.388) and placebo groups (triangles, slope -0.262).

For the planned Phase II trial of PB in combination with TUDCA, we therefore selected a dose of 1 gram of TUDCA twice a day (2 grams per day) as a target dose.

Ursodiol (UDCA), the non-taurine conjugated form of TUDCA, was also found to be safe and well-tolerated in a crossover study subjects with ALS<sup>18</sup>. Subjects who received UDCA treatment also showed significant benefit as measured by the Appel ALS rating scale.

AMX-0035 in ALS

Protocol Number: AMX3500


Subjects randomized to active therapy in the Phase II trial will receive 3g PB and 1g TUDCA twice a day orally (or by feeding tube). AMX0035 will be presented as a 4 gram sachet to be suspended in water and taken with a glass of water before a meal. Single agent TUDCA or PB treatment in subjects with ALS was very well tolerated.

In the TUDCA study from Elia et al., the AE profile and laboratory anomalies were not different between the TUDCA and placebo cohort. In the small group of 15 subjects treated with TUDCA, the adverse events were limited to diarrhea.

In the PB study from Cudkowicz et al., tolerability was similar to that reported in other trials of PB in other indications. There were no changes in safety laboratory tests, EKG or vital signs. The most common AEs were those previously reported with PB, including falls, dizziness, diarrhea, edema, dry mouth, headache, nausea and rash. A single subject interrupted treatment with PB at the 9 gram per day dose (i.e. a dose higher than that planned in the proposed Phase II) for the occurrence of edema on the foot and under the eye.

## 2.1.4 Additional Previous Clinical Experience with Phenylbutyrate

Sodium phenylbutyrate (PB) is generally well tolerated. It is FDA approved for subjects with urea cycle disorders including deficiencies of carbamylphosphate synthetase, ornithine transcarbamylase, or argininosuccinic acid synthetase. It is indicated in patients with either neonatal-onset deficiency or late-onset disease. The usual total daily dose is 450-600 mg/kg/day in patients weighing less than 20kg, or 9.9-13.0 g/m<sup>2</sup>/day in larger patients. Detailed information can be found on the package insert for PB<sup>19</sup>.

Sodium phenylbutyrate is also under development as an anticancer agent. In a dose escalation study in subjects with refractory solid tumor malignancies doses of up to 45g/day were administered<sup>20</sup>. Due to dose-limiting toxicities, the study concluded that 27g/day was the maximally tolerated dose. Nausea, vomiting, hypocalcemia and fatigue occurred at the 36g/day and 45g/day doses. Gastrointestinal upset (nausea, dyspepsia and vomiting) occurred at the lowest dose of 9g/day and was seen within 30 minutes of drug ingestion. However, 82% of subjects completed the study despite these side effects. Other frequently reported side effects include a "sweat"-like odor, usually noticeable only to the caregiver. Mild neurotoxicity (confusion, lethargy) has been noted at higher doses of close to 30g/day, but resolved with dose reduction.

A dose-escalation study of intravenous PB in subjects with myelodysplastic syndromes and acute myelogenous leukemia found a maximally tolerated dose at 375 mg/kg/day (26.3g/day for a 70kg individual) with no serious toxicities detected in subjects receiving doses between 125 and 375 mg/kg/day (8.8 and 26.3g/day for a 70kg individual) <sup>21</sup>. Dose-limiting toxicities (lethargy, confusion, slurred speech) were detected at 440 and 500 mg/kg/day PB (30.8 and 35g/day respectively, for a 70kg individual). Reports of edema have been blamed on the high sodium

AMX-0035 in ALS Protocol Number: AMX3500


load associated with the drug. Phase I/II studies in subjects with sickle cell anemia (see table 1 below) and beta thalassemia report similar side effects.

Another phase I study in subjects with refractory solid tumors tested IV PB doses between 150 to 515 mg/kg/day (up to 36g/day for a 70kg individual) with dose-limiting toxicities (excessive somnolence, confusion) and electrolyte abnormalities resulting at a dose of 515 mg/kg/day (36.0 g/day for a 70kg individual). The maximally tolerated dose of PB was determined to be 410 mg/kg/day (28.7 grams/day for a 70kg individual) as there were no dose-limiting toxicities at this dose and no subjects required dose reductions or escalations (see table 1).

The most common side effects of PB include: menstrual irregularities, decreased appetite, sweat-like body odor, and bad taste. Less common side effects include: nausea, vomiting, stomach upset, stomach pain, gastritis, headache, and skin rash. Rarely, cases of peptic ulcers, rectal bleeding, constipation, pancreatitis and renal tubular acidosis have been reported. Hypoalbuminemia, metabolic acidosis, alkalosis, hyperchloremia, hyperuricemia, hypokalemia, hypophosphatemia, hyperphosphatemia and hypernatremia have been observed. At higher doses, some subjects experienced confusion and fatigue, both of which resolved with dose reductions. Rarely, the following may occur, but have not been directly linked to sodium phenylbutyrate therapy: anemia, leukopenia, leukocytosis, thrombocytopenia, thrombocytosis, arrhythmia, syncope and depression.

**Table 1: Prior Clinical Experience with Phenylbutyrate** 

| Dose | Durati | Patient | # of | AE summary | Location | Status | Reference | NCT # (if ref |
|---|---|---|---|---|---|---|---|---|
| | on | Population | patients | | | | | unavailable) |
| 9-21g/day | | | | | | | | |
| | 5 | Amyotrophic | 40 | Well tolerated at | US | Completed | Amyotrophic | |
| | months | Lateral | | 9 g | | | Lateral | |
| | | Sclerosis | | | | | Sclerosis. | |
| | | | | | | | 2009; 10: | |
| | | | | | | | 99106 | |
| 12-18g/day | | | | | | | | |
| | 28 days | Huntington's | 24 | Table included, | US | Completed | Hogarth et al. | |
| | per | | | Nausea, | | | Sodium | |
| | dose | | | Headache, gain | | | phenylbutyrat | |
| | level | | | instability, were | | | e in | |
| | | | | most common. | | | Huntington's | |
| | | | | Most side effects | | | disease: a | |
| | | | | uncommon at | | | dose-finding | |
| | | | | 12g/day | | | study. Mov. | |
| | | | | | | | Disord. 2007. | |
| 15g/day | | | | | | | | |
| | 12 | SCA3 | 20 | NA | Ex-US | Withdrawn | NA | NCT01096095 |
| | months | | | | | | | |
| 500mg/kg/day | | | | | | | | |
| | 14 days | Maple Syrup | 40 | NA | US | Complete | Brunetti-Pieri, | NCT01529060 |
| | | Urine Disease | | | | | et al. | |

AMX-0035 in ALS

Protocol Number: AMX3500


| Dose | Durati<br>on | Patient<br>Population | # of patients | AE summary | Location | Status | Reference | NCT # (if ref<br>unavailable) |
|---|---|---|---|---|---|---|---|---|
| | | | | | | | Phenylbutyrat<br>e therapy for<br>maple syrup<br>urine disease.<br>Hum. Mol.<br>Gen. 2010. | |
| 20g/day | 4 days | Urea Cycle<br>Disorders | 9 | NA | US | Active | NA | NCT02111200 |
| IV<br>Phenylbutyrate | 7 years | Advanced<br>Colorectal<br>Cancer | 46 | NA | US | Cancelled | NA | NCT00002796 |
| 12.4g/day<br>(mean dose,<br>198mg/kg-<br>476mg/kg<br>range) | 12<br>months | Urea Cycle<br>Disorders | 11 | One case of<br>vomiting, see<br>horizon package<br>insert | US | Completed | Lichter-<br>Konecki, U. et<br>al. Mol Genet<br>Metab. 2011<br>Aug;103(4) | |
| <20g/day | 10<br>weeks | Urea Cycle<br>Disorders | 14 | See Horizon package insert | US | Completed | See Horizon<br>Package Insert | |
| 1g/day | 16<br>weeks | HIV | 279 | NA | Ex-US | Completed | NA | NCT01702974 |
| 9-36g/day | 28 days | recurrent<br>malignant<br>glioma | 23 | No AE's at<br>9g/day, 1<br>headache, 1<br>lightheadedness<br>at 18g/day, 1<br>fatigue at<br>27g/day, 2<br>fatigue at<br>36g/day | US | Completed | Neuro-oncol.<br>2005 Apr | |
| 1g/day | 16<br>weeks | Tuberculosis | 390 | NA | Ex-US | Completed | BMC<br>Pulmonary<br>MedicineBM<br>C series 2013 | |
| Effective dose for UCD | 28 days | UCD | 46 | 1 patient<br>experienced<br>Hyperammonaem<br>ia | US | Completed | NA | NCT00992459 |
| 450-<br>600mg/kg/day | 18-24<br>months | SMA | 14<br>infants | NA | US | Completed | NA | NCT00528268 |
| 19g p.o./day<br>divided into<br>three doses | 1 week | F(del)508 CF | 18 | Minimal and comparable side effects | US | Completed | Am J Respir<br>Crit Care<br>Med. 1998 | |

Protocol Number: AMX3500


| Dose | Durati<br>on | Patient<br>Population | # of patients | AE summary | Location | Status | Reference | NCT # (if ref<br>unavailable) |
|---|---|---|---|---|---|---|---|---|
| 500mg/kg/day | 12<br>weeks | SMA1 | 5 | Terminated for slow enrollment | US | Cancelled | NA | NCT00439218 |
| 500mg/kg/day | 12<br>weeks | SMA2/SMA3 | 9 | Terminated for poor compliance | US | Cancelled | NA | NCT00439569 |
| 500mg/kg/day | 1 week | Argininosucci<br>nic Aciduria | 12 | NA | US | Completed | NA | NCT00345605 |
| 200mg/kg IV | 5 days | Acute<br>Myeloid<br>Leukemia | 10 | Well tolerated,<br>fatigue observed | US | Completed | Leukemia (20<br>06) 20, 212–<br>217 | |
| 7.5g/day | 2<br>weeks | BMI>27 | 10 | NA | Canada | Completed | NA | NCT00533559 |
| IV<br>Phenylbutyrate | NA | Multiple<br>Cancers | 20 | NA | US | Completed | NA | NCT00006019 |
| IV<br>Phenylbutyrate | up to<br>4yrs | AML | 9 to 24 | NA | US | Completed | NA | NCT00006240 |
| IV/Oral<br>Phenylbutyrate<br>Escalating top<br>dose: 45g/day | 4<br>weeks | Refractory<br>Solid Tumor<br>malignancies | 28 | Generally well<br>tolerated<br><27g/day.<br>Nausea,<br>Hypocalemia<br>observed | US | Completed | Clin Cancer<br>Res August<br>2001 7;2292 | |
| 7.5g, 15g/day | 14 day | Protinuric<br>Nephropathy | 26 | NA | Ex-US | Completed | NA | NCT02343094 |
| IV<br>Phenylbutyrate | Ascend ing Dose | Hematologic<br>Cancer | 3 to 24 | NA | US | Completed | NA | NCT00006239 |
| 20g/day | 41 to<br>460<br>days | Thalessemia<br>Major | 11 | Weight gain and/or edema caused by increase salt load in 2/12, transient epigastric discomfort in 7/12, and abnormal body odor in 3/12 subjects | US | Completed | AF Collins et<br>al., 1995;<br>Blood: 85 (1) | |

Protocol Number: AMX3500


| Dose | Durati | Patient | # of | AE summary | Location | Status | Reference | NCT # (if ref |
|---|---|---|---|---|---|---|---|---|
| | on | Population | patients | | | | | unavailable) |
| 20g/day | 41 to | Thalessemia | 11 | Weight gain | US | Completed | January 1, | |
| | 460 | Major | | and/or edema | | | 1995; Blood: | |
| | days | | | caused by | | | 85 (1) | |
| | | | | increase salt load | | | | |
| | | | | in 2/12, transient | | | | |
| | | | | epigastric | | | | |
| | | | | discomfort in | | | | |
| | | | | 7/12, and | | | | |
| | | | | abnormal body | | | | |
| | | | | odor in 3/12 | | | | |
| | | | | subjects | | | | |
| 20g/day | 4 | Healthy, BMI | 101 | Not yet posted | US | Completed | NA | NCT00771901 |
| | weeks | 30-45 | | | | | | |
| 30-40g/day | 10 days | ATT | 12 | NA | US | Completed | NA | NCT00067756 |
| | | deficiency | | | | | | |

### 2.1.5 Additional Previous Clinical Experience with TUDCA

Tauroursodeoxycholic acid is currently marketed in Italy under the brand name Tudcabil ( ). It is exported to China and Turkey under the brand name Taurolite. It is used for the treatment of cholesterol gallstones. It has been used for the treatment of cholestatic liver diseases including primary cirrhosis, pediatric familial intrahepatic cholestasis and primary sclerosing cholangitis and cholestasis due to cystic fibrosis. To our knowledge there are no other off label uses of tauroursodeoxycholic acid.

Ursodeoxycholic acid (UDCA), which is widely used in the United States for treating gallstones, is produced and secreted endogenously by the liver as a taurine (TUDCA) or glycine (GUDCA) conjugate. Taurine conjugation increases the solubility of UDCA by making it more hydrophilic. TUDCA is taken up in the distal ileum under active transport and therefore likely has a slightly a longer dwell time within the intestine than UDCA which is taken up more proximally in the ileum (IND

TUDCA is widely used for the dissolution of cholesterol gallstones. This generally requires long periods of treatment often 1 to 2 years to obtain complete dissolution (IND ).

Between 1997 and 2007, 898,000 Tudcabil tablets were sold in Italy (taken from product profile contained in referenced IND \_\_\_\_\_\_\_). There were no reported cases of toxicity related to Tudcabil capsules. There were no reports of overdose or drug abuse during this period. There were no reports related to the use of pregnancy (all pregnant subjects, and those planning to become pregnant, are excluded from this trial). Common adverse events include mild abdominal pain and diarrhea. There are some cases of pruritus and a very limited number of cases of elevated liver enzymes. It should be noted that most of the studies are conducted in subjects with chronic liver disease.

AMX-0035 in ALS Protocol Number: AMX3500


TUDCA is contraindicated in subjects with biliary tree infections, frequent biliary colic, or in subjects who have trouble absorbing bile acids (e.g. ileal disease or resection). The only known or theoretical drug interactions are with substances that inhibit the absorption of bile acids such as cholestyramine and with drugs that increase the elimination of cholesterol in the bile (TUDCA reduces biliary cholesterol content). Based on similar physicochemical characteristics, it is likely that drug toxicity and interactions are very similar to those of ursodeoxycholic acid which are summarized below.

TUDCA has been and is being evaluated in multiple other studies as well. A study at Columbia of 20 subjects with new onset type 1 diabetes in which subjects are administered 1.75g TUDCA for 12 months is ongoing (see table 2). A study at Washington University assessing the effect of TUDCA on lipid markers and ER stress has been completed in 101 subjects at 1.75g daily for 4 weeks; an additional study arm in this study assessed PB at 20g/day (see table 2). We have included in the IND package a signed right to reference to the IND for a study at Washington University assessing subjects with HIV receiving 1.75g daily TUDCA for 30 days.

Table 2: Prior Clinical Experience with TUDCA

| TUDC | Duration | Patient Exp | # of | AE summary | Location | Status | Reference | NCT# |
|---|---|---|---|---|---|---|---|---|
| A Dose | | Population | patients | , | | | | |
| 1g b.i.d. | | 1. | 1,000 | | | | | |
| | 1 year | Amyotrophic<br>Lateral<br>Sclerosis | 29 | Mild diarrhea occurred in two patients treated with TUDCA and in two treated with placebo; anorexia was reported in a placebo-treated patient. | ex-US | Complete d | Elia et al.<br>European J.<br>Neurology | NCT00877604 |
| 1.75g/d<br>ay | 1 year | Type 1 Diabetes | 20 | NA | US | Ongoing | NA | NCT02218619 |
| 1.75g/d<br>ay | 4 weeks | Healthy, BMI<br>30-45 | 101 | Not yet posted | US | Complete d | NA | NCT00771901 |
| 750mg/<br>day | 24 weeks | Chronic<br>Cholestatic<br>Liver Disease | 199 | NA | Ex-US | Complete d | NA | NCT01829698 |
| 750mg/<br>day | 18<br>months | Transthyretin<br>Amyloid<br>Cardiomyopath<br>y | 40 | NA | US | Active | NA | NCT01855360 |
| 1.75g<br>once | 30 days | Protease- | 48 | NA | US | Recruiting | NA | NCT01877551 |

AMX-0035 in ALS

Protocol Number: AMX3500


| TUDC<br>A Dose | Duration | Patient<br>Population | # of patients | AE summary | Location | Status | Reference | NCT# |
|---|---|---|---|---|---|---|---|---|
| daily | | inhibitor<br>Associated<br>Insulin<br>Resistance | | | | | | |
| 750mg/<br>day | 12<br>months | PBC | 216 | NA | Ex-US | Complete d | NA | NCT01857284 |
| 750mg/<br>day | 1 year | Transthyretin<br>Amyloidosis | 40 | NA | Ex-US | Complete d | NA | NCT01171859 |
| UNK | 3 months | Hepatobiliary<br>Disease in<br>Cystic Fibrosis | 39 | NA | US | Complete d | NA | NCT00004441 |
| 500mg/<br>day | 60-80<br>days | Biliary<br>Dyspepsia | 30 | Safe and well tolerated | Ex-US | Complete<br>d | Rivista di<br>Patologia e<br>Clinica, 1985,<br>34:3370-380 | |
| 750mg/<br>day | 254 days<br>mean | Cholelithiasis | 93 | Minor side effects<br>were observed in 4<br>patients treated with<br>TUDCA (2 g.i. and 2<br>unspecified skin<br>cases) none of which<br>required suspension<br>of treatment. | Ex-US | Complete d | Acta Toxicologica et Therapeutica, Vol. 5, Oct- Dec. 1986, Vaccari ed., Parma | |
| 1.0<br>g/day | 10 days | Patients with<br>Gallstones | 7 | NA | US | Complete<br>d | Batta, et al.<br>Hepatology,<br>1982, 2(6):811-<br>816 | |
| .5g, 1g,<br>1.5g/da<br>y | 6 months | Primary Biliary<br>Cirrhosis | 24 | Diahrrea only<br>observed AE | Ex-US | Complete d | Crosignani, et<br>al. Digestive<br>Diseases and<br>Sciences. 1996,<br>41(4):809-815 | |
| .5g, 1g,<br>1.5g/da<br>y | 6 months | Primary Biliary<br>Cirrhosis | 24 | NA | Ex-US | Complete d | Setchell et al.<br>GUT, 1996;<br>38:439-446 | |
| 3.5-<br>16.6mg<br>/kg/day | 4-6 weeks | Gallstones | 33 | NA | Ex-US | Complete d | Muraca et al. International J. Clin. Pharmacol. Therapeutices, 1995; 33(7):391-393, | |

Protocol Number: AMX3500


| TUDC<br>A Dose | Duration | Patient<br>Population | # of<br>patients | AE summary | Location | Status | Reference | NCT# |
|---|---|---|---|---|---|---|---|---|
| 3.5-<br>16.6mg<br>/kg/day | 4-6 weeks | Biliary Lipid<br>Composition | 33 | NA | Ex-US | Complete d | Muraca et al.<br>Ital J.<br>Gastroenterol<br>1995, 27:439-<br>440 | |
| 10mg/k<br>g/day | 1 month | Gallstones | 29 | NA | Ex-US | Complete d | Portincasa, et<br>al. Ital. J.<br>Gastroenterol.<br>1996, 28:111-<br>113 | |
| 10-<br>13mg/k<br>g/day | 3 months | chronic hepatitis | 5 | NA | Ex-US | Complete d | Panella, et al.<br>Ital. J.<br>Gastroenterolog<br>y 1995; 27:256-<br>258; | |
| 10mg/k<br>g/day | 6 months | Gallstones | 12 | No side effects<br>observed | Ex-US | Complete d | La Clinica<br>Terapeutica,<br>1986; 117:475-<br>479 | |
| 10mg/k<br>g/day | 6 months | Gallstones | 31 | NA | Ex-US | Complete d | The American<br>Journal of<br>Gastroenterolog<br>y 1995;<br>90(6):978-981 | |
| 500mg/<br>day | 3 months | Biliary<br>Dyspepsia | 133 | NA | Ex-US | Complete d | Advances in<br>Therapy - 1994;<br>11 (1):34-41, | |
| 500mg/<br>day | 3 months | chronic active<br>hepatitis | 53 | No side effects<br>observed | Ex-US | Complete<br>d | Portincasa et al.<br>Current<br>Therapeutic<br>Research. 1993;<br>53(5):521-531 | |
| 500mg/<br>day | 3 months | Patients post<br>cholecystectom<br>y | 203 | 1 patient vomited,<br>and 1 had abdominal<br>pain in active, 1<br>abdominal pain, 1<br>rash cutaneous, 1<br>lipotinemia in<br>placebo | Ex-US | Complete d | Annali Italiani<br>di Chirurgia,<br>1993,<br>64(5):533-537 | |
| .5g, 1g,<br>1.5g/da<br>y | 6 months | asymptomatic/m<br>ildly<br>symptomatic<br>PBC | 24 | NA | Ex-US | Complete d | Hepatology, 1994, 130A. | |

Protocol Number: AMX3500


| TUDC<br>A Dose | Duration | Patient<br>Population | # of<br>patients | AE summary | Location | Status | Reference | NCT # |
|---|---|---|---|---|---|---|---|---|
| .5g, 1g,<br>1.5g/da<br>y | 6 months | asymptomatic/m<br>ildly<br>symptomatic<br>PBC | 24 | TUDCA was well<br>tolerated (rarely<br>diarrhoea dose<br>dependent<br>reversible). | Ex-US | Complete d | Hepatology,<br>1993, 10; 176A | |
| 500mg/<br>day | 6 months | PBC | 23 | Well tolerated and<br>no patient<br>complained of side<br>effects. | Ex-US | Complete<br>d | Aliment. Pharmacol. Ther. 1997; 11:409-414 | |
| 750mg/<br>day | 2 month<br>with<br>crossover | PBC | 12<br>females | NA | US | Complete d | Hepatology.<br>1999; 29:320-<br>327 | |
| 675mg/<br>day | 2 months | PBC | 15 | Two patients experienced burning discomfort in the epigastrium during the TUDCA treatment period. | Ex-US | Complete d | Clin. Res. 1986,<br>34(1):181 | |
| 13mg/k<br>g/day | 3 months | Chronic liver<br>disease<br>hystologically<br>determined | 69 | NA | Ex-US | Complete d | J of<br>Hepatology.<br>1993; 18<br>(Suppl. 1) S157 | |
| 500mg/<br>day | 3 months | chronic hepatitis | 134 | 2.2% cases of<br>diarrhoea solved<br>promptly without<br>suspension of<br>therapy | Ex-US | Complete d | Advances in therapy. 1994, 11(5):262-268 | |
| 500mg/<br>day | 3 months | patients with<br>biopsy proved<br>CAH due to<br>HCV or HBV<br>infections | 162 | 1 patient developed<br>abdominal<br>discomfort, 1 patient<br>had mild pruritus, 3<br>patients developed<br>mild diarrhoea<br>without wirthdrawal | Ex-US | Complete d | Current<br>Therapeutic<br>Research 1995;<br>56(6):626-634, | |
| 500mg/<br>day | 6 months | compensated<br>liver cirrhosis<br>associated with<br>hepatitis B or C<br>of Child's group<br>A or B<br>(histological<br>tests) | 30 | No side effects and<br>no treatment<br>withdrawals<br>occurred | Ex-US | Complete d | Current<br>Therapeutic<br>Research 1994;<br>55 (11):1355-<br>1362, | |

Protocol Number: AMX3500


| TUDC<br>A Dose | Duration | Patient<br>Population | # of<br>patients | AE summary | Location | Status | Reference | NCT # |
|---|---|---|---|---|---|---|---|---|
| Phase | | 1 opulation | patients | | | | | |
| Phase 1: TUDC A 10 mg/kg/ day + lympho blastoid IFNa 3MU/m 2 ter in week; Phase 2: TUDC A idem + IFNa tapering dose down to the minimu m effectiv e | 6 month<br>phase 1, 6<br>months<br>phase 2 | Patients with CHC | 120 | NA | Ex-US | Complete | Gastroenterolog<br>y 1996; 110(4)<br>A1296. | |
| .25, .5,<br>1 g/day | 6 months | Chronic<br>Hepatitis | 155 | Two patients were withdrawn for minor side effects (one for diarrhea and one for dyspepsia). | Ex-US | Complete d | Hepatology.<br>1995,<br>23(4):120A - 53 | |
| 500mg/<br>day | 12<br>months | Liver transplant | 33 | Safe and well<br>tolerated | Ex-US | Complete d | Ital J. Gastro<br>and Hepatology<br>1999; P/C<br>13/37:154 | |

### 2.1.6 Previous Clinical Experience with Ursodiol (UDCA)

Ursodiol therapy has not been associated with liver damage. Lithocholic acid, a naturally occurring bile acid, is known to be a liver-toxic metabolite. This bile acid is formed in the gut from ursodiol less efficiently and in smaller amounts than that seen from chenodiol. Lithocholic acid is detoxified in the liver by sulfation and, although man appears to be an efficient sulfater, it is possible that some subjects may have a congenital or acquired deficiency in sulfation, thereby predisposing them to lithocholate-induced liver damage (IND

Abnormalities in liver enzymes have not been associated with Actigall® (Ursodiol USP capsules) therapy and, in fact, Actigall® has been shown to decrease liver enzyme levels in liver disease. However, subjects given Actigall® should have SGOT (AST) and SGPT (ALT)

AMX-0035 in ALS

Protocol Number: AMX3500


measured at the initiation of therapy and thereafter as indicated by the particular clinical circumstances.

Bile acid sequestering agents such as cholestyramine and colestipol may interfere with the action of ursodiol by reducing its absorption. Aluminum-based antacids have been shown to adsorb bile acids in vitro and may be expected to interfere with ursodiol in the same manner as the bile acid sequestering agents (IND \_\_\_\_\_\_\_). Estrogens, oral contraceptives, and clofibrate (and perhaps other lipid-lowering drugs) increase hepatic cholesterol secretion, and encourage cholesterol gallstone formation and hence may counteract the effectiveness of ursodiol.

Ursodeoxycholic acid was tested in 2-year oral carcinogenicity studies in CD-1 mice and Sprague-Dawley rats at daily doses of 50, 250, and 1000 mg/kg/day. It was not tumorigenic in mice. In the rat study, it produced statistically significant dose-related increased incidences of pheochromocytomas of adrenal medulla in males (p=0.014, Peto trend test) and females (p=0.004, Peto trend test). A 78-week rat study employing intrarectal instillation of lithocholic acid and tauro-deoxycholic acid, metabolites of ursodiol and chenodiol, has been conducted. These bile acids alone did not produce any tumors. A tumor-promoting effect of both metabolites was observed when they were co-administered with a carcinogenic agent. Ursodiol is not mutagenic in the Ames test (IND

#### 2.2 Potential Risks and Benefits

#### 2.2.1 Potential Risks

The safety profile with PB administration is in large part derived from studies of subjects with urea cycle disorders. Refer to the phenylbutyrate tablet label (Buphenyl®).

In female subjects, the most common clinical adverse event reported was amenorrhea/menstrual dysfunction (irregular menstrual cycles), which occurred in 23% of the menstruating subjects. Decreased appetite occurred in 4% of all subjects. Body odor (probably caused by the metabolite, phenylacetate [PAA]) and bad taste or taste aversion were each reported in 3% of subjects.

AMX-0035 in ALS Protocol Number: AMX3500


Other adverse events reported in 2% or fewer subjects were:

- Gastrointestinal: abdominal pain, gastritis, nausea and vomiting; constipation, rectal bleeding, peptic ulcer disease, and pancreatitis each occurred in one subject.
- Hematologic: aplastic anemia and ecchymoses each occurred in one subject.
- Cardiovascular: arrhythmia and edema each occurred in one subject.

• Renal: renal tubular acidosis

• Psychiatric: depression

• Skin: rash

• Miscellaneous: headache, syncope, and weight gain

Phenylbutyrate has been evaluated in a dose-escalating study in ALS subjects over the course of 20-weeks and was found to be generally safe and tolerable<sup>15</sup>. Specifically, the most common adverse events included falls or other accidental injury, dizziness, diarrhea, edema, dry mouth, headache, nausea, and rash. With the exception of headache, these adverse events occurred at a higher rate compared to the comparison placebo cohort. These events are expected side effects from PB. There were no clinically significant changes in laboratory values, EKGs or vital signs. No deaths or unexpected and related serious adverse events occurred. Significant adverse events did not occur more frequently with subjects who were taking riluzole in addition to NPB, compared to subjects taking PB alone. Importantly, this study evaluated daily dosages of phenylbutyrate between 9 and 21 grams while our study will be limited to 6 grams daily.

Neurotoxicity was reported in cancer subjects receiving intravenous phenylacetate, 250–300 mg/kg/day for 14 days, repeated at 4-week intervals. Manifestations were predominately somnolence, fatigue, and lightheadedness; with less frequent headache, dysgeusia, hypoacusis, disorientation, impaired memory, and exacerbation of a pre-existing neuropathy.

These adverse events were mainly mild in severity. The acute onset and reversibility when the phenylacetate infusion was discontinued suggest a drug effect.

The most common adverse reactions reported with the use of TUDCA (≥1%) are: abdominal discomfort, abdominal pain, diarrhea, nausea, pruritus, and rash.

TUDCA is generally well tolerated. A derivative, UDCA or ursodiol, is approved for subjects with primary biliary cirrhosis. Common adverse events with TUDCA include mild abdominal pain and diarrhea. There are some cases of pruritus and a very limited number of cases of elevated liver enzymes.

TUDCA has been evaluated over a year-long placebo controlled study in ALS subjects at 1g b.i.d<sup>17</sup>. The population for safety analysis consisted of 15 subjects who took TUDCA and 14 subjects who took placebo. The treatment was well tolerated in all subjects. Laboratory parameters did not change in either treatment group during the course of the study. Except for

AMX-0035 in ALS

Protocol Number: AMX3500


the expected complications related to ALS, no changes in vital signs and laboratory values that could possibly be attributed to the study drug or placebo were recorded. Overall, five adverse events were considered by the Investigators to be study related based on the subjects' descriptions. Two events were reported in the 15 TUDCA-treated subjects (13.3%); three events occurred in the 14 placebo-treated subjects (21.4%). The events were as follows: mild diarrhea occurred in two subjects treated with TUDCA and in two treated with placebo; anorexia was reported in a placebo-treated subject. Four subjects died during the study period, one in the TUDCA group and three in the placebo group. The one death in the treated group was not considered drug related—TUDCA trended towards a survival benefit.

The risks and side effects of muscle strength testing include fatigue and/or muscle cramping.

#### 2.2.2 Known Potential Benefits

This study is designed to assess the safety, tolerability and biological activity of AMX0035 therapy. TUDCA and PB have both been tested individually in ALS clinical trials and met their primary endpoints of safety and tolerability. TUDCA also met its efficacy endpoint of slowing ALSFRS-R decline, and PB was therapeutically efficient in improving histone acetylation levels. If successful, this trial will allow further clinical development of this therapy to potentially slow ALS progression. The trial is also assessing multiple biomarkers in concert with clinical endpoints, which will allow both a more detailed understanding of drug activity as well as serve as a data set for the field as a whole to help understand how these biomarkers might track ALS progression.


#### **3 OBJECTIVES**

### 3.1 Study Objectives

This Phase II protocol is intended as a proof of concept of AMX0035 as a safe and effective treatment of adult subjects with ALS. The main strategic objectives of this protocol are below.

The primary outcome measures will be:

- 1. To confirm the safety and tolerability of a fixed-dose combination of PB and TUDCA in subjects with ALS over a 6-month period;
- 2. To measure the impact of the treatment using the slope of progression with the revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R);

The secondary objectives of the study will be:

- 1. To assess the impact of AMX0035 on the rate of decline of isometric muscle strength, as measured by the Accurate Test of Limb Isometric Strength (ATLIS);
- 2. To assess the impact of AMX0035 on disease progression as measured by Slow Vital Capacity (SVC) decline, time to tracheostomy and survival;
- 3. To assess the impact of AMX0035 on biomarkers including phosphorylated axonal neurofilament H subunit (pNF-H) levels and 18 kDa translocator protein (TSPO) uptake;
- 4. To develop concentration-response models of TUDCA and phenylbutyrate at steady-state after administration of AMX0035 sachet twice-daily.
- 5. To measure the impact of AMX0035 on survival.

## 3.2 Study Outcome Measures

## 3.2.1 Primary Outcome Measures

The primary outcome measures for the study will include:

- Safety and tolerability as defined as the proportion of subjects able to remain on study drug until planned discontinuation.
- The rate of decline (slope of decline) in the ALS functional rating scale (ALSFRS-R).

Safety and tolerability will be assessed by the procedures outlined in Section 9.

The revised version of the ALSFRS was created to add assessments of respiratory dysfunction, including dyspnea, orthopnea, and the need for ventilatory support. The revised ALSFRS (ALSFRS-R) has been demonstrated to retain the properties of the original scale and show strong internal consistency and construct validity.

Survival endpoint will be defined as death, tracheostomy or permanent assisted ventilation (>22 hours a day).

AMX-0035 in ALS Protocol Number: AMX3500


### 3.2.2 Secondary Outcome Measures

The secondary outcome measures include:

- Assessing the impact of AMX0035 on the rate of decline of isometric muscle strength, as measured by the Accurate Test of Limb Isometric Strength (ATLIS);
- Assessing the impact of AMX0035 on disease progression as measured by Slow Vital Capacity (SVC) decline;
- Assessing the impact of AMX0035 on survival, hospitalization and tracheostomies;
- Assessing the impact of AMX0035 on biomarkers including phosphorylated axonal neurofilament H subunit (pNF-H) levels and 18 kDa translocator protein (TSPO) uptake;
- Assessing the concentration-response model of TUDCA and phenylbutyrate at steady-state after administration of AMX0035 4 grams twice daily.


## 4 STUDY DESIGN

### 4.1 Overall Study Design and Plan

During the enrollment period approximately 176 subjects will be screened from approximately 25 Northeast ALS Consortium (NEALS) centers in the US. One hundred thirty-two (132) of these subjects will be randomly assigned in a 2:1 ratio to oral (or feeding tube) twice daily sachet of active therapy or matching placebo. Treatment duration will be twenty-four (24) weeks. For the first three weeks study drug will be administered once daily. If tolerated, the dose will then be increased to twice a day. Clinic visits will occur at Screening, Baseline, Week 3 (day 21), Week 6 (day 42), Week 12 (day 84), Week 18 (Day 126), and Week 24 (Day 168). Phone calls will be conducted at Week 9, Week 15, Week 21 and Week 28 (4 weeks after completion of treatment).

All visit windows are consecutive calendar days and are calculated from the day the subject starts study treatment (Day 0, the day of the Baseline Visit). Any change from this visit window will be considered an out of window visit deviation.

An one thirty-two (132) week Open Label Extension (OLE) study will be available to those subjects who complete the randomized, double-blind study. Please refer to 13.7 Appendix VII for all the details on the OLE.

#### 4.2 Study Centers

This study will be conducted at up to 25 NEALS Centers in the US. Sites will be selected based on recruitment record from prior trials, compliance with prior study protocols and regulations, clinical research expertise and availability of necessary resources.

#### 4.3 Study Duration

Subjects will remain on randomized, placebo-controlled, double-blind treatment until the Week 24 visit. Each randomized subject will also have a Follow-up Telephone Interview 28 days after the completion of dosing to assess for adverse events (AEs), changes in concomitant medications and to administer the ALSFRS-R. Including the Screening and Follow-up Visits, each subject will be in the study for approximately 8 months. We expect the study to take up to 18 months to meet enrollment goals.

#### 4.4 Protocol Adherence

Each Site Investigator must adhere to the protocol detailed in this document and agree that any changes to the protocol must be approved by the NCRI Coordination Center (CC) or their Central Institutional Review Board (cIRB). Each Site Investigator (SI) will be responsible for enrolling only those study subjects who have met protocol eligibility criteria.

AMX-0035 in ALS Protocol Number: AMX3500

### 5 STUDY ENROLLMENT AND WITHDRAWAL

## 5.1 Number of Study Subjects

Approximately 132 ALS subjects will be randomized.

#### 5.2 Inclusion and Exclusion Criteria

#### 5.2.1 Inclusion Criteria

Inclusion Criteria

- 1. Male or female, aged 18-80 years of age
- 2. Sporadic or familial ALS diagnosed as definite as defined by the World Federation of Neurology revised El Escorial criteria
- 3. Less than or equal to 18 months since ALS symptom onset
- 4. Capable of providing informed consent and following trial procedures
- 5. Geographically accessible to the site
- 6. Slow Vital Capacity (SVC) >60% of predicted value for gender, height, and age at the Screening Visit
- 7. Subjects must either not take riluzole or be on a stable dose of riluzole for at least 30 days prior to the Screening Visit. Riluzole-naïve subjects are permitted in the study.
- 8. Women of child bearing potential (e.g. not post-menopausal for at least one year or surgically sterile) must agree to use adequate birth control for the duration of the study and 3 months after last dose of study drug
  - a. Women must not be planning to become pregnant for the duration of the study and 3 months after last dose of study drug
- 9. Men must agree to practice contraception for the duration of the study and 3 months after last dose of study drug
  - a. Men must not plan to father a child or provide sperm for donation for the duration of the study and 3 months after last dose of study drug

Acceptable birth control methods for use in this study are:

- Hormonal methods, such as birth control pills, patches, injections, vaginal ring, or implants
- Barrier methods (such as a condom or diaphragm) used with a spermicide (a foam, cream, or gel that kills sperm)
- Intrauterine device (IUD)
- Abstinence (no heterosexual sex)
- Unique partner who is surgically sterile (men) or not of child bearing potential (female)

**Date of ALS Symptom Onset.** For the purposes of this study, the date of symptom onset will be defined as the date the subject first had symptoms of their disease, i.e., weakness. To be eligible

AMX-0035 in ALS Protocol Number: AMX3500


for this study, the date of symptom onset must be no greater than exactly 18 months prior to the Screening Visit date.

### **MR-PET Sub-Study**

A subset of study subjects will undergo MR-PET and will need to meet the following additional inclusion criteria:

- 1. Ability to safely lie flat for 90 min for MR-PET procedures in the opinion of the Site Investigator
- 2. High or mixed affinity to bind TSPO protein (Genotype Ala/Ala or Ala/Thr)

**TSPO affinity test:** Venous blood for the TSPO affinity test will be drawn from all subjects who have indicated their interest in participating in the MR-PET sub-study. (This will be indicated via a checkbox on the consent form.) The blood will be drawn at Screening in order to have the subjects genotyped for the Ala147Thr TSPO polymorphism in the *TSPO* gene (rs6971). About 10% of humans show low binding affinity to PBR28<sup>21</sup>.

**Note:** High or Mixed affinity binders (Ala/Ala or Ala/Thr) will be considered eligible, whereas the low affinity binders (Thr/Thr) will be considered ineligible for the MR-PET sub-study.

**Note:** A subject may be eligible for the main study but ineligible for the MR-PET sub-study. However, if a subject is found to be ineligible for the main study, he or she is automatically ineligible for the MR-PET sub-study as well.

#### **5.2.2** Exclusion Criteria

Study subjects meeting any of the following criteria during screening evaluations will be excluded from entry into the study:

#### **Exclusion Criteria**

- 1. Presence of tracheostomy
- 2. Exposure to PB, TUDCA or UDCA within 3 months prior to the Screening Visit or planning to use these medications during the course of the study
- 3. History of known allergy to PB or bile salts
- 4. Abnormal liver function defined as AST and/or ALT > 3 times the upper limit of the normal
- 5. Renal insufficiency as defined by eGFR < 60 mL/min/1.73m<sup>2</sup>.
- 6. Poorly controlled arterial hypertension (SBP>160mmHg or DBP>100mmHg) at the Screening Visit
- 7. Pregnant women or women currently breastfeeding
- 8. History of cholecystectomy

AMX-0035 in ALS Protocol Number: AMX3500


- 9. Biliary disease which impedes biliary flow including active cholecystitis, primary biliary cirrhosis, sclerosing cholangitis, gallbladder cancer, gallbladder polyps, gangrene of the gallbladder, abscess of the gallbladder.
- 10. History of Class III/IV heart failure (per New York Heart Association NYHA)
- 11. Severe pancreatic or intestinal disorders that may alter the enterohepatic circulation and absorption of TUDCA including biliary infections, pancreatitis and ileal resection
- 12. The presence of unstable psychiatric disease, cognitive impairment, dementia or substance abuse that would impair ability of the subject to provide informed consent, according to Site Investigator judgment
- 13. Patients who have cancer with the exception of the following: basal cell carcinoma or successfully treated squamous cell carcinoma of the skin; cervical carcinoma in situ; prostatic carcinoma in situ; or other malignancies curatively treated and with no evidence of disease recurrence for at least 3 years.
- 14. Clinically significant unstable medical condition (other than ALS) that would pose a risk to the subject if they were to participate in the study
- 15. Active participation in an ALS clinical trial evaluating an experimental small molecule within 30 days of the Screening Visit. (*Please refer to MOP section E.* Protocol Compliance for current list of experimental small molecules).
- 16. Exposure at any time to any cell therapies and gene therapies under investigation for the treatment of subjects with ALS (off-label use or investigational)
- 17. Exposure to monoclonal antibodies under investigation for the treatment of ALS (off-label use or investigational) within 90 days from screening. If previously exposed to monoclonal antibodies under investigation for the treatment of ALS, a 90-day wash-out period will be required prior to screening.
- 18. Implantation of Diaphragm Pacing System (DPS)
- 19. Anything that, in the opinion of the Site Investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study
- 20. Exposure to any disallowed medications listed below

### **MR-PET Sub-Study**

A subset of study subjects will undergo MR-PET. The following additional exclusion criteria apply to this subset:

- 1. Exposure to immunomodulatory medications within 30 days of the Screening
- 2. Any contraindication to undergo MRI studies such as:
  - a. History of a cardiac pacemaker or pacemaker wires
  - Metallic particles in the body
  - c. Vascular clips in the head
  - Prosthetic heart valves
  - e. Severe claustrophobia impeding ability to participate in an imaging study

AMX-0035 in ALS Protocol Number: AMX3500


- 3. Low affinity binders (Thr/Thr) on the TSPO Affinity Test
- 4. Radiation exposure that exceeds the site's current guidelines

**Note:** A subject may be eligible for the main study but ineligible for the MR-PET sub-study. However, if a subject is found to be ineligible for the main study, he or she is automatically ineligible for the MR-PET sub-study as well.

**Note on Benzodiazepines for MR-PET Sub-Study Subjects:** If an MR-PET subject is taking a benzodiazepine, he or she should not take the benzodiazepine for at least 1 day before his or her scans with the exception of lorazepam and clonazepam that do not need to be discontinued.

## Disallowed medications for all subjects include

- HDAC Inhibitors including:
  - Valproate
  - Vorinostat (Zolinza)
  - o Romidepsin
  - o Chidamide
  - o Panobinostat
  - o Lithium
  - o Butyrate
  - o Suramin
- Probenecid
- Bile Acid Sequestrants including:
  - o Cholestyramine and Cholestyramine Light
  - Questran and Questran Light
  - o Welchol
  - Colestid and Colestid Flavored
  - o Prevalite

## Note on Antacids Within Two Hours of AMX0035 Administration:

Antacids containing Aluminum hydroxide or smectite (aluminum oxide) may not be taken within two hours of administration of AMX0035 as they inhibit absorption of TUDCA. These include:

- o Alamag
- o Alumina and Magnesia
- o Antacid, Antacid M and Antacid Suspension
- o Gen-Alox
- Kudrox
- o M.A.H.

AMX-0035 in ALS

Protocol Number: AMX3500

 $Version\ 7.0$ 

- Maalox HRF and Maalox TC
- Magnalox
- Madroxal
- o Mylanta and Mylanta Ultimate
- o Ri-Mox
- o Rulox

## **Cautionary Note on Mexiletine**

Subjects who participated in the Mexiletine trial within the last 30 days will be excluded from the trial. However, subjects who are using Mexiletine at a dosage less than or equal to 300mg/day for cramps and fasciculations will not be excluded.

There is a potential for an interaction between AMX0035 and Mexiletine; at 20 times the intended clinical concentration (C<sub>max</sub>), the principal metabolite of Phenylbutyrate, Phenylacetylacetate has been shown to be inhibitory to CYP 1A2 and CYP 2D6 which are the major enzymes responsible for the breakdown of Mexiletine. Therefore, it is possible the co-administration of Phenylbutyrate and Mexiletine will increase the subject's exposure to Mexiletine.

Subjects who are co-administered AMX0035 and Mexiletine should therefore be monitored for Mexiletine-associated adverse events, and if these events present, the Site Investigator should consider stopping or reducing the dosage of Mexiletine. Adverse events associated with Mexiletine include but are not limited to cardiac arrhythmias, liver injury, and blood dyscrasias.

## **5.3** Treatment Assignment Procedures

Each subject who meets all eligibility criteria will be randomized to receive either therapy by twice daily sachet of AMX0035 (3g PB and 1g TUDCA) or matching placebo for 24 weeks of treatment. For the first three weeks of the study subjects will only take a single sachet daily and will be instructed to increase to 2 sachets daily at the Week 3 Visit.

### 5.3.1 Randomization Procedures

The randomization scheme will be independently developed and will indicate the treatment assignment and the subject numbers to be used by each site. The randomization scheme will be managed by the manufacturer.

### 5.4. Reasons for Withdrawal

A study subject will be discontinued from participation in the study if:

- Any clinical adverse event (AE), laboratory abnormality, requirement for a concomitant medication, concurrent illness, or other medical condition or situation occurs such that, in the opinion of the Investigator, continued participation in the study would not be in the best interest of the subject.
- The subject is non-compliant or is lost-to-follow-up.

AMX-0035 in ALS

Protocol Number: AMX3500


Subjects are free to withdraw from participation in the study at any time upon request.

## **5.4.1** Handling of Withdrawals

A subject may choose to discontinue participation in the study at any time. However, the Site Investigator (SI) or designee will encourage subjects to continue with follow-up, regardless of their compliance with the study drug. If the SI or designee is concerned about the use of a prohibited medication or other safety issues, then the study drug may have to be reduced to single dose or discontinued. If a subject permanently discontinues study drug, the SI or designee should still encourage subjects to follow the study protocol under the modified intent-to-treat principle (ITT). These subjects will be encouraged to follow the study visits, off drug. Loss to follow-up should be prevented whenever possible.

Any subject who is on study drug and needs to begin the use of any prohibited medication, must immediately discontinue use of the study drug and should not begin use of the prohibited medication before an appropriate wash-out period of at least 30 days occurs. Subjects who must permanently discontinue study drug may continue in the ITT portion of the study, per protocol.

Subjects who permanently discontinue study drug and will not continue monitoring per the study schedule should complete early study drug termination procedures per protocol. Subjects who discontinue treatment should not be unblinded unless there is a specific reason to do so.

If a subject wishes to withdraw consent, i.e., withdraw his or her participation in future study procedures, the subject will be asked to delay consent withdrawal to allow for a Final Safety Visit and Final Safety Telephone Call. The subject will be asked to return to the study site for a Final Safety Visit as soon as possible after stopping study drug, if possible within 28 days of asking to withdraw consent. The subject will also be asked to have a Follow-Up Telephone Call no sooner than 28 days (+5 days) after taking their last dose of study drug to monitor their safety and to permit review of their medical records at the end of the study to document their vital status.

Subjects who withdraw from the study due to adverse events will be followed for outcome measures under the ITT protocol as noted above. The DSMB will review these events promptly and make recommendations about potential changes to the study, including possible changes to protocol, updates to the informed consent form, or even ending the study early.

In the event a subject wishes to no longer have their personal health information used for the analysis of this study, he or she will notify the site through an authorized letter and future data will not be included in analysis; however, all data up to this letter will still be included.

AMX-0035 in ALS Protocol Number: AMX3500


## 5.5 Termination of Study

This study may be prematurely terminated if, in the opinion of the DSMB or sponsor, there is sufficient reasonable cause. Written notification, documenting the reason for study termination, will be provided to the Principal Investigator or Sponsor by the terminating party.

Circumstances that may warrant termination include, but are not limited to:

- Determination of unexpected, significant, or unacceptable risk to subjects.
- Enrollment is unsatisfactory.
- Insufficient adherence to protocol requirements.
- Data that are not sufficiently complete and/or evaluable.
- Plans to modify, suspend or discontinue the development of the study drug.

If the study is prematurely terminated or suspended, the Sponsor will promptly inform the Site Investigators/institutions, and the regulatory authority(ies) of the termination or suspension and the reason(s) for the termination or suspension. The Central IRB (cIRB) will also be informed promptly and provided the reason(s) for the termination or suspension by the Sponsor or by the Site Investigator/institution, as specified by the applicable regulatory requirement(s).

#### 6 TREATMENTS ADMINISTERED

#### **6.1** Treatments

## **6.1.1 Study Product Description**

AMX0035 is a combination therapy comprised of two active pharmaceutical ingredients, sodium phenylbutyrate (PB and tauroursodeoxycholic acid (TUDCA).

Phenylbutyrate is an approved compound in the United States for urea cycle disorders and is marketed in the US as Buphenyl<sup>®</sup>. There is an existing USP monograph for this material. The chemical structure for PB is provided below.

## **Chemical Structure PB**

The drug substance PB is produced by conditions. The manufacture and controls for PBA are described in Drug Master File No.

The specifications for PB are identical to those of the Ph.Eur.

The drug substance TUDCA is currently marketed in Italy under the brand name Tudcabil. It is exported to China and Turkey under the brand name Taurolite. It is used for the indications of treatment of cholesterol gallstones. It has been used for the treatment of cholestatic liver diseases including primary cirrhosis, pediatric familial intrahepatic cholestasis and primary sclerosing cholangitis and cholestasis due to cystic fibrosis. To our knowledge, there are no other uses of tauroursodeoxycholic acid. It is marketed by some companies in the United States on websites such as Amazon as a dietary supplement to "promote liver health".

The chemical structure for TUDCA is provided below.

AMX-0035 in ALS Protocol Number: AMX3500




The drug substance TUDCA is produced by

The specifications for TUDCA are identical to those used by the supplier.

A powder filled sachet will be used as the AMX0035 drug product. The drug product will be filled under cGMP conditions in an aluminum foil lined sachet.

The sachet containing active ingredients will include:

- o Active Ingredients:
  - 1g TUDCA
  - 3g PB
- o Excipients
  - Sodium Phosphate Dibasic, Anhydrous
  - Dextrates, Hydrates
  - Sorbitol
  - Syloid 63FP (colloidal silica)
  - Sucralose
  - Sodium Stearyl Fumarate
  - Weber Mixed Berry Flavoring
  - Kleptose Linecaps (maltodextrin)

### 6.1.2 Placebo

A matched placebo will be used to maintain the dosage-blind. The placebo sachets for this study will match the corresponding AMX0035 sachets in size, color, and presentation.

The placebo sachets contain:

- Excipients
  - Sodium Phosphate Dibasic, Anhydrous
  - Dextrates, Hydrates

AMX-0035 in ALS

Protocol Number: AMX3500


- Sorbitol
- Syloid 63FP (colloidal silica)
- Sucralose
- Sodium Stearyl Fumarate
- Weber Mixed Berry Flavoring
- Kleptose Linecaps (maltodextrin)
- Denatonium Benzoate Granules

Administration of matching placebo will be the same as for subjects in the treatment group.

## 6.2 Acquisition

Upon receipt of the study treatment supplies, an inventory must be performed and a drug receipt log filled out and signed by the person accepting the shipment. It is important that the designated study staff counts and verifies that the shipment contains all the items noted in the shipment inventory. Any damaged or unusable study drug in a given shipment will be documented in the study files. The Site Investigator must notify the study Sponsor or their designee of any damaged or unusable study treatments that were supplied to the Site Investigator's site.

## 6.2.1 Formulation, Packaging, and Labeling

The study drug is prepackaged in kits containing 98 sachets and ready for oral (or feeding tube) administration. The Site Investigator (SI) has the responsibility to ensure that the integrity of packaged study drug is not jeopardized prior to dispensing. Each individual subject kit must be dispensed as provided with no further repackaging or labeling done at the investigational site, unless required by the institution per institutional polices.

### **6.2.2** Product Storage and Stability

The SI must ensure that all investigational drug supplies are kept in a locked, safe area at ambient temperature 15-25°C with access limited to authorized study staff. Investigational drug supplies should not be repackaged in any way.

Once subjects have access to kits containing the sachets, they will be asked to store them away from moisture at room temperature. Stability has been assessed both at ICH standard and accelerated conditions for each of the individual active ingredients and they were found to be stable over five years. Drug product will receive regular stability testing over the course of the study to ensure product does not degrade. At least one month stability will be verified prior to initiation of the proposed trial. Subjects should contact the SI or their designee in the case of damaged goods; the SI or designee will coordinate with the Sponsor or their designee to determine the most appropriate remediation.

### **6.2.3 Dispensing Product**

Drug product will be dispensed to subjects only after the SI has reviewed the necessary safety procedures for the subject to continue taking the study drug. Safety procedures must be

AMX-0035 in ALS Protocol Number: AMX3500


performed every six (6) months to monitor safety. Interim safety procedures can be done at each study visit, at the discretion of the SI.

Drug product can be dispensed from the site to the subject using the following options:

- 1. The drug product will be dispensed to the subject at the clinic visit.
- 2. The drug product will be delivered to the subject's home of residence through the use of a clinical supply chain courier company.
- 3. Other options may be approved by the Sponsor on an ad hoc basis.

# 6.3 Dosage, Preparation and Administration of Study Intervention/Investigational Product

It is recommended that the study drug be taken prior to a meal. Subjects should rip open the sachet of study drug and add it to a cup or other container and add approximately 8 oz. (1 cup) of room temperature water and stir vigorously. The study drug mixture should be consumed completely and within one hour of combining the contents of the sachet with water. The site personnel will provide oral instructions to the patients and will assist the patient through the first oral administration (Appendix VI).

Subjects may resume normal eating and drinking after taking the study drug.

## **Note on Antacids Within Two Hours of Study Drug Administration**

Antacids containing Aluminum hydroxide or smectite (aluminum oxide) may not be taken within two hours of administration of the study drug as they inhibit absorption of TUDCA.

These include:

- o Alamag
- o Alumina and Magnesia
- o Antacid, Antacid M and Antacid Suspension
- o Gen-Alox
- o Kudrox
- o M.A.H.
- Maalox HRF and Maalox TC
- Magnalox
- Madroxal
- Mylanta and Mylanta Ultimate
- o Ri-Mox

AMX-0035 in ALS

Protocol Number: AMX3500

 $Version\ 7.0$ 

#### $\circ$ Rulox

## **6.3.1** Feeding Tube Study Drug Administration

For subjects with a gastrostomy or nasogastric (feeding) tube, the study drug may be dissolved in water as per the procedures outlined above in Section 6.3 and the study drug may be administered via the feeding tube.

## 6.4 Modification of Study Intervention/Investigational Product For A Subject

Any dosage adjustment, including the reason for and dates of adjustment, will be documented in the CRF for each subject requiring this manipulation. The SI or designated licensed physician Sub-Investigator may reduce the dosage of study drug or discontinue the study drug in its entirety for adverse events (AEs) thought to be related to the study drug or for other reasons during the trial (the reason for, and dates of suspension or dose reduction must be documented). All dose modifications need to be discussed with the study Medical Monitor. If the AE is mild or moderate, the dosage may be reduced until the event improves. The SI or designated licensed physician Sub-Investigator may then choose to resume the higher dosage or maintain the subject at a reduced dosage.

If the event is serious or life threatening, and deemed to be definitely drug related, the study drug will be discontinued immediately. Study subjects must remain off the study drug permanently. Subjects may not resume study drug. All AEs will be followed to resolution within the study for 28 days (+ 5 days) after a subject's last dose of study drug.

## **6.4.1.** Dosage Discontinuation

Reasons for discontinuation of study drug may include an AE, Medical Monitor or Site Investigator recommendation, Sponsor termination, protocol deviation, lost-to-follow-up, subject request, or death. All serious adverse events (SAEs) that occur in a subject who has discontinued early must be recorded and reported within 24-hours of awareness.

Study subjects who discontinue study drug prematurely (early termination from study) and decide to not remain in the modified intent-to-treat (ITT) portion of the study will be encouraged to return for a Final Safety/Early Termination Visit and participate in a Follow-Up Telephone Call 28 days (+ 5 days) after the last dose of study drug.

All subjects who discontinue study drug early and choose to remain in the ITT portion of the study will be encouraged to follow the study visits, off drug, up to the time of the last visit (Follow-Up Telephone Call).

SAEs will be followed for resolution for 28 days (+5 days) after a subject's last dose of study drug, regardless of whether they prematurely discontinued study drug or completed 24 weeks of treatment.

AMX-0035 in ALS Protocol Number: AMX3500


## 6.5 Study Drug Accountability Procedures

At the completion of the study, there will be a final reconciliation of study drug shipped, drug consumed, and drug remaining. This reconciliation will be logged on the study drug reconciliation form, signed and dated. Any discrepancies noted will be investigated, resolved, and documented prior to return or destruction of unused study drug. Drug destroyed on site will be documented in the study files.

## 6.6 Assessment of Subject Compliance

Subjects will be instructed to return empty and unused study drug containers at each clinic Visit (Weeks 6, 12, 18, and 24) or the Final Safety Visit (whichever occurs first). In the event that a remote study visit occurs, the subject will be instructed to return empty and unused study drug containers from previous study drug kits at the next clinic visit.

Site staff will count returned and unused sachets to determine compliance.

Non-compliance will be otherwise defined as taking less than 80% or more than 125% of study drug as determined by sachet counts. If a study subject is non-compliant with study drug, the Site Investigator (SI) or designee should re-educate and train the subject in administration of study drug. Data indicating non-compliance will be used in the end of study analysis.

## 6.7 Prior and Concomitant Therapy

Throughout the study, Site Investigators (SIs) may prescribe concomitant medications or treatments deemed necessary to provide adequate supportive care provided that the medications are licensed in the United States. Study subjects should not receive other experimental agents during the study. This includes marketed agents at experimental dosages that are being tested for the treatment of ALS. All concomitant medications and/or treatments and significant non-drug therapies including supplements and assistive devices, received by a subject should be recorded on the appropriate source document and eCRF.

Any investigational small molecule therapy being used or evaluated for the treatment of ALS is prohibited beginning 30 days prior to the Screening Visit and throughout the study. This includes, but is not limited to, the following:

- Pioglitazone
- Arimoclomol
- Olanzapine
- Tamoxifen
- NP001
- Mexiletine
- Rasagiline
- Masitinib
- Dexpramipexole
- Tirasemtiv

AMX-0035 in ALS

Protocol Number: AMX3500


- Ibudilast
- TW001
- Inosine
- RNS60
- Acetyl-L-Carnitine
- Methylcobalamine (if administered at doses equal to or greater than 25 mg per week)

Use of any biologic therapy prior to this study excludes subjects from enrollment. This includes any cell or gene therapy under evaluation for the treatment of ALS and includes but is not limited to, the following:

- ISIS 333611
- Ionis SOD1R
- NurOwn
- Q-Cells
- NSI-566
- GM604
- GSK 1223249
- Treg cell therapies

### 6.7.1 Prohibited Medications and Contraindications

### **Prohibited Medications**

Throughout the course of the trial, study subjects should not be treated with the following medications. If a Site Investigator learns that a subject has begun therapy with any of these medications, this should be reported to the Medical Monitor and Coordination Center immediately and the SI should make the determination whether to stop the study drug or the prohibited medication immediately, taking into account the health, safety and preference of the study subject.

Agents which might impair bile acid processing or renal function are contraindicated with AMX0035. Prohibited medications include but are not limited to:

- HDAC Inhibitors including:
  - o Valproate
  - Vorinostat (Zolinza)
  - o Romidepsin
  - o Chidamide
  - Panobinostat
  - o Lithium

AMX-0035 in ALS

Protocol Number: AMX3500


- o Butyrate
- o Suramin
- Probenecid for potential kidney interaction
- Antacids containing aluminum hydroxide or smectite (aluminum oxide) within two hours of administration of AMX0035. These inhibit absorption of TUDCA. These include:
  - Alamag
  - o Alumina and Magnesia
  - o Antacid, Antacid M and Antacid Suspension
  - o Gen-Alox
  - Kudrox
  - o M.A.H.
  - o Maalox HRF and Maalox TC
  - Magnalox
  - Madroxal
  - Mylanta and Mylanta Ultimate
  - o Ri-Mox
  - o Rulox
- Bile Acid Sequestrants including:
  - o Cholestyramine and Cholestyramine Light
  - Questran and Questran Light
  - Welchol
  - Colestid and Colestid Flavored
  - o Prevalite

## **Pregnancy & Nursing Mothers**

There are no adequate and well-controlled studies in pregnant women. <u>Female subjects or female partners of male subjects should not become pregnant during the study or 3 months after stopping study drug.</u>

If a female subject becomes pregnant, study treatment must be discontinued immediately. If a female subject becomes pregnant during the course of the study, the Medical Monitor and Coordination Center should be contacted immediately.

It is not known whether AMX0035 is excreted in human milk. Caution should be exercised; therefore, no subject should nurse an infant while participating in this study.

AMX-0035 in ALS Protocol Number: AMX3500


## 7 STUDY SCHEDULE

No study procedures should be performed prior to the signing of the informed consent form (ICF). All subjects will sign an ICF prior to undergoing any study tests or procedures. It is recommended that the ALSFRS-R be completed first at every visit. After the ALSFRS-R it is recommended that SVC and ATLIS measurements are performed so as not to fatigue the subject with other testing. Blood samples are recommended to be taken at the end of the study visits. The order of testing, however, will be at the discretion of each Site Investigator (SI).

Visit windows are consecutive calendar days and the target visit dates are calculated from the Baseline Visit.

Subjects who withdraw consent or early terminate from the study (i.e., discontinue study drug) will be asked to come in for a Final Safety Visit and have a Final Follow-up Telephone Call 28 days (+5 days) after stopping study drug.

## 7.1 MR-PET Scheduling Call

Subjects from all sites will be considered to participate in the MR-PET Sub-Study. The MR-PET Sub-Study procedures will be conducted at Massachusetts General Hospital (MGH) in Boston, MA. However, blood will be drawn for TSPO testing at the subject's site during the Screening Visit.

Subjects participating in the MR-PET Sub-Study may be consented over the phone by a medically licensed professional MGH study staff member to determine subject eligibility and to ensure the subject is safe to undergo the MR-PET scan. These procedures include:

- Obtain verbal pre-screening informed consent from subject
- o Assess MR-PET inclusion and exclusion criteria
- o Complete MR-PET safety questionnaire

During this call, MR-PET Sub-Study procedures will be discussed in detail and the subject should be given the opportunity to ask questions about the MR-PET Sub-Study. The MGH study staff will write a consent note to document the consenting process over the phone. The written informed consent will be signed by the subject and the MGH Study Investigator at the MR-PET in-person visit.

## 7.2 Screening Visit

The following procedures will be performed at an office visit to determine the subject's eligibility for the study.

- Obtain written informed consent from subject
- o Create Globally Unique Identifier (GUID)
- Assess inclusion and exclusion criteria
- Obtain medical history and demographics
- o Review and document concomitant medications and therapies

AMX-0035 in ALS

Protocol Number: AMX3500


- Obtain ALS diagnosis history
- o Administer ALSFRS-R questionnaire
- o Perform pulmonary function testing including slow vital capacity (SVC)
- o Measure isometric strength using ATLIS machine
- o Assess and document adverse events (AEs) that occur after subject signs informed consent form (ICF)
- o Measure vital signs (blood pressure, heart and breathing rates, temperature)
- o Perform neurological examination
- o Perform comprehensive physical examination including height and weight
- o Perform 12-lead ECG (Electrocardiogram)
- [After other tests] Collect blood samples for clinical laboratory assessments including Hematology (CBC with differential), Complete Chemistry Panel, Liver Function Tests, and serum pregnancy test (for women of child-bearing potential [WOCBP])
- o MR-PET SCAN SUBJECTS ONLY: TSPO Affinity Testing
- o Collect urine sample for urinalysis
- Schedule the Baseline Visit

**MR-PET Scan:** For those subjects that consent to participate in the MR-PET scan sub-study, the scan will be scheduled/performed <u>before</u> the Baseline Visit at the MGH in Boston, MA. At that time, blood will also be collected for peripheral blood mononuclear cell (PBMC) storage and analysis.

#### 7.2.1 Screen Failures

Any subject who signs consent will be considered enrolled in the study. If a subject fails screening, at a minimum, the following information should be captured and entered in the Electronic Data Capture (EDC) System:

- o Inclusion/Exclusion Criteria
- Demographics
- o Reason for screen failure

## 7.3 MR-PET Visit 1 (Only for patients in MR-PET substudy)

The following procedures will be performed at an office visit to determine the subject's eligibility for the MR-PET sub-study.

- Obtain written informed consent
- o Assess MR-PET inclusion and exclusion criteria
- o Complete MR-PET safety questionnaire
- o Perform the MR-PET Scan
- o Perform the Upper Motor Neuron-Burden (UMN-B) Scale
- o Measure vital signs (blood pressure, heart and breathing rates, temperature), and weight
- o Administer ALSFRS-R questionnaire
- Collect blood for
  - o Biomarker (PBMC) testing

AMX-0035 in ALS

Protocol Number: AMX3500


- o Pregnancy testing (for women of child bearing potential)
- o Review and document concomitant medications and therapies
- Assess and document adverse events (AEs) that occur after subject signs informed consent form (ICF)

## **MR-PET Follow-Up Call**

This visit will take place 24-48 hours after the MR-PET Visit 1. The following procedures will be performed.

Assess and document AEs directly related to the MR-PET procedures

#### 7.4 Baseline Visit

This visit will take place a maximum of 42 days after the Screening Visit. The 42-day window allows those subjects participating in the MR-PET portion of the study to have their scans scheduled. Site staff are advised to schedule the baseline visit as soon as possible after determining eligibility. The following procedures will be performed.

- o Confirm eligibility criteria are still met
- o Randomize subject using kit number from the study drug
- o Administer the C-SSRS baseline questionnaire
- o Administer ALSFRS-R questionnaire
- o Perform pulmonary function testing, including slow vital capacity (SVC)
- o Measure isometric strength using ATLIS machine
- o Review and document concomitant medications and therapies
- Review and document Adverse Events since last visit and following study drug administration
- Measure vital signs
- o [After other tests] Collect blood samples for clinical laboratory assessments including Hematology (CBC with differential), Complete Chemistry Panel, Liver Function Tests.
- Collect blood sample for biomarkers
- o Collect pre-dose blood sample for pharmacokinetic analysis
- Collect blood sample for optional DNA collection (Note: if Baseline visit has passed or blood sample for DNA was not collected, the blood sample should be collected at the next available visit)
- o Collect urine sample for urinalysis

After all other visit activities are completed:

- o Dispense 6 weeks of study drug
- o Administer first dose of study drug. The healthcare staff member will advise the subject on appropriate administration (Appendix VI). The subject will be observed at the site for a minimum of 60 minutes by an appropriate healthcare staff member according to the

AMX-0035 in ALS Protocol Number: AMX3500


- site's institutional/state regulations to assess medical status and any immediate reaction to the study drug.
- o Review and document any Adverse Events after first dose of study drug

### 7.5 Week 3 Clinic Visit

This visit will take place 21±5 days after the Baseline Visit. The following procedures will be performed.

- o Administer ALSFRS-R questionnaire
- o Review and document concomitant medications and therapies
- Review and assess Adverse Events
- o Measure vital signs
- o Administer the C-SSRS questionnaire
- Collect blood samples for clinical laboratory assessments including Hematology (CBC with differential), Complete Chemistry Panel, Liver Function Tests
- o Collect urine sample for urinalysis
- o Perform study drug accountability
- o Unless drug is not tolerated, advise subject to increase dosage level from one sachet to two sachets daily.
- Schedule next study visit

#### 7.6 Week 6 Clinic Visit

This visit will take place 42±5 days after the Baseline Visit. The following procedures will be performed.

- o Administer ALSFRS-R questionnaire
- o Perform pulmonary function testing, including slow vital capacity (SVC)
- o Measure isometric strength using ATLIS machine
- o Review and document concomitant medications and therapies
- o Review and assess Adverse Events
- Measure vital signs
- o Administer the C-SSRS questionnaire
- o [After other tests] Collect blood samples for clinical laboratory assessments including Hematology (CBC with differential), Complete Chemistry Panel, Liver Function Tests
- Collect blood sample for biomarkers
- o Collect urine sample for urinalysis
- o Perform study drug accountability and collect all unused study drug and empty containers
- o Dispense next 6 weeks of study drug
- Schedule next study visit

## 7.7 Week 9 Telephone Visit

This visit will take place 63±5 days after the Baseline Visit. The following procedures will be performed.

o Administer ALSFRS-R questionnaire

AMX-0035 in ALS

Protocol Number: AMX3500

 $Version\ 7.0$ 

- Review and document concomitant medications and therapies
- Assess and document AEs
- Enquire about tolerance and compliance
- o Schedule next study visit
- o Remind subject to bring study drug to the Week 12 Visit

## 7.8 Week 12 Clinic Visit

This visit will take place 84±5 days after the Baseline Visit. Subject must take study drug at the site upon beginning this visit due to the PK analysis. It is recommended that this visit happens earlier in the day since the drug is administered in clinic. The following procedures will be performed:

- o Record day/time of previous study drug dose, including if the subject missed a dose.
- Note time of last meal
- o Administer study drug and record time of administration
- o Collect blood sample for PK (i.e. at 1-hour or 4-hours post-dose) as indicated at the time of randomization
- Administer ALSFRS-R questionnaire
- o Perform pulmonary function testing including slow vital capacity (SVC)
- o Measure isometric strength using ATLIS machine
- o Review and document concomitant medications and therapies
- Review and assess Adverse Events
- o Measure vital signs
- o Perform neurological examination
- o Perform comprehensive physical examination including weight
- o Perform 12-lead ECG (Electrocardiogram)
- o Administer the C-SSRS questionnaire
- o [After other tests] Collect blood samples for clinical laboratory assessments including Hematology (CBC with differential), Complete Chemistry Panel, Liver Function Tests
- Collect blood sample for biomarkers
- o Collect urine sample for urinalysis
- o Perform study drug accountability and collect all unused study drug and empty containers
- o Dispense next 6 weeks of study drug
- Schedule next study visit

## 7.9 Week 15 Phone Visit

This visit will take place 105±5 days after the Baseline Visit. The following procedures will be performed.

- Administer ALSFRS-R questionnaire
- o Review and document concomitant medications and therapies
- Assess and document AEs
- o Enquire about tolerance and compliance
- Schedule next study visit

AMX-0035 in ALS

Protocol Number: AMX3500


#### 7.10 Week 18 Clinic Visit

This visit will take place 126±5 days after the Baseline Visit. The following procedures will be performed.

- Administer ALSFRS-R questionnaire
- o Perform pulmonary function testing including slow vital capacity (SVC)
- o Measure isometric strength using ATLIS machine
- o Review and document concomitant medications and therapies
- Review and assess Adverse Events
- Measure vital signs
- o Administer the C-SSRS questionnaire
- o [After other tests] Collect blood samples for clinical laboratory assessments including Hematology (CBC with differential), Complete Chemistry Panel, Liver Function Tests
- Collect blood sample for biomarkers
- Collect urine sample for urinalysis
- o Perform study drug accountability and collect all unused study drug and empty containers
- o Dispense next 6 weeks of study drug
- Schedule next study visit

#### 7.11 Week 21 Phone Visit

This visit will take place 147±5 days after the Baseline Visit. The following procedures will be performed.

- Administer ALSFRS-R questionnaire
- o Review and document concomitant medications and therapies
- Assess and document AEs
- o Enquire about tolerance and compliance
- o Schedule next study visit
- o Remind subject to bring study drug to clinic for the Week 24 Visit
- Schedule MR-PET scan for those subjects participating in the MR-PET Sub-Study

## 7.12 MR-PET Visit 2 (Only for patients in MR-PET Substudy)

This visit will take place between the Week 12 and Week 20 study visits.

- Complete MR-PET safety questionnaire
- o Perform the MR-PET Scan
- o Perform the Upper Motor Neuron-Burden (UMN-B) Scale
- o Measure vital signs (blood pressure, heart and breathing rates, temperature), height, and weight
- o Administer ALSFRS-R questionnaire
- Collect blood for
  - o Biomarker (PBMC) testing
  - o Pregnancy testing (for women of child bearing potential)

AMX-0035 in ALS

Protocol Number: AMX3500


- Review and document concomitant medications and therapies
- Assess and document adverse events (AEs)

## MR-PET Follow-Up Call

This visit will take place 24-48 hours after the MR-PET Visit 2. The following procedures will be performed.

o Assess and document AEs directly related to the MR-PET procedures

## 7.13 Final Study Visit (Week 24)

This visit will take place 168±5 days after the Baseline Visit. Subject must take study drug upon beginning this visit due to the PK analysis. It is recommended that this visit happens earlier in the day since the drug is administered in clinic. The following procedures will be performed:

- o Record day/time of previous study drug dose, including if the subject missed a dose
- o Record time of last meal
- o Administer study drug and record time of administration
- o Collect a single blood sample for PK (i.e. at 1 hour or 4 hours post-dose) as indicated at the time of randomization (Week 24 only, not Early Termination Subjects)
- o Administer ALSFRS-R questionnaire
- o Perform pulmonary function testing, including slow vital capacity (SVC)
- o Measure isometric strength using ATLIS machine
- o Review and document concomitant medications and therapies
- o Review Adverse Events
- o Measure vital signs
- o Perform neurological examination
- o Perform physical examination including weight
- o Perform 12-lead ECG (Electrocardiogram)
- o Administer the C-SSRS questionnaire
- o Exit questionnaire
- [After other tests] Collect blood samples for clinical laboratory assessments including Hematology (CBC with differential), Complete Chemistry Panel, Liver Function Tests
- Collect blood sample for biomarkers
- o Collect urine sample for urinalysis
- o Perform study drug accountability and collect all unused study drug and empty containers

### 7.14 Final Follow-up Telephone Call (Week 28)

A follow-up phone call will take place 28 + 5 days (no earlier than 28 days) after the subject's last dose of study drug. Subjects who enroll in the open label extension will not be required to complete this telephone call. The following will be performed.

- o Complete ALSFRS-R Questionnaire
- o Review and document concomitant medications and therapies
- Assess and document AEs

AMX-0035 in ALS

Protocol Number: AMX3500


## 7.15 Withdrawal of Consent Final Safety Visit & Final Follow-up Telephone Call

Subjects who withdraw consent will be asked to come in for a Final Safety Visit as soon as possible after consent withdrawal and to have a final Follow-Up Telephone Call 28 + 5 days (no earlier than 28 days) after the last dose of study drug.

The following will be performed at the Final Safety Visit:

- o Administer ALSFRS-R questionnaire
- o Perform pulmonary function testing, including slow vital capacity (SVC)
- o Measure isometric strength using ATLIS machine
- o Review and document concomitant medications and therapies
- o Review Adverse Events
- Measure vital signs
- o Perform physical examination including weight
- o Perform neurological examination
- o Perform 12-lead ECG (Electrocardiogram)
- o Administer the C-SSRS questionnaire
- o [After other tests] Collect blood samples for clinical laboratory assessments including Hematology (CBC with differential), Complete Chemistry Panel, Liver Function Tests
- Collect blood sample for biomarkers
- o Collect urine sample for urinalysis
- o Perform study drug accountability and collect all unused study drug and empty containers

The following procedures will be performed via telephone 28 +5 days after the last administration of study drug:

- o Administer ALSFRS-R questionnaire
- o Review and document concomitant medications and therapies
- Assess and document AEs

#### 7.16 Protocol Deviations

A protocol deviation is any noncompliance with the clinical trial protocol. The noncompliance may be either on the part of the subject, the Site Investigator, or the study site staff. As a result of deviations, corrective actions are to be developed by the site and implemented promptly.

All deviations from the protocol must be addressed in the subject's source documents. All major protocol deviations will be sent to the central IRB and entered in the Protocol Deviations Log in the Electronic Data Capture (EDC) System.

### 7.16.1 Missed Visits and Procedures

Missed visits and any procedures not performed (not attempted) for reasons other than illness, injury or progressive disability (i.e. subject is physically unable to perform test) will be reported as protocol deviations.

AMX-0035 in ALS Protocol Number: AMX3500


Procedures or visits not performed due to illness, injury or disability, including procedures that were attempted but failed (i.e. blood samples unable to be drawn after multiple attempts, or weight unable to be obtained due to subject immobility) will not be reported as protocol deviations.

Study drug compliance that is outside the limits set in the study operations manual will be reported as a protocol deviation.

In the event that a remote study visit occurs, the following procedures should be completed in the suggested order: ALSFRS-R, AE Review, Key Study Events, Concomitant Medications, Columbia-Suicide Severity Scale. Missed procedures during these remote visits will not be considered protocol deviations.

Details and specific instructions regarding protocol deviations, including any exceptions to this standard procedure, are found in the Site Manual of Procedures.

## 7.17 Recording Deaths

Information on whether a subject has died may be obtained by the subject's family, clinic notes, or utilizing public means such as a reliable internet source such as the Centers for Disease Control and Prevention (CDC) National Death Index (http://www.cdc.gov/nchs/ndi.htm) or the Social Security Death Index (http://ssdmf.info/).

#### 8 CLINICAL ASSESSMENTS AND OUTCOME MEASURES

#### 8.1 Clinical Variables

Assessments will be performed at designated time-points throughout the study for clinical evaluation. In addition to the assessments evaluated below, subjects will provide information on their demographics, past medical history, including ALS and cardiac history, as well as concomitant medication usage.

## 8.1.1 Vital Signs, Height & Weight

Vital signs will be obtained after the subject has been in a seated position for several minutes. Vital signs, including systolic and diastolic blood pressure, pulse rate (radial artery)/minute, respiratory rate/minute, temperature and weight will be assessed at specified visits. Height will be measured and recorded at the Screening Visit only.

## **8.1.2** Clinical Laboratory Assessments

The following laboratory tests will be performed for safety:

- Hematology with differential panel: complete blood count with differential (hematocrit, hemoglobin, platelet count, RBC indices, Total RBC, Total WBC, and WBC & differential)
- O Blood chemistry panel/Liver function tests (LFTs): alanine aminotransferase (ALT (SGPT)), aspartate aminotransferase (AST (SGOT)), albumin, alkaline phosphatase, bicarbonate, blood urea nitrogen, calcium, chloride, creatinine, glucose, magnesium, phosphate, potassium, sodium, total bilirubin and total protein
- O Urinalysis: albumin, bilirubin, blood, clarity, color, glucose, ketones, nitrate, pH, protein, specific gravity, urobilinogen and WBC screen
- Serum human chorionic gonadotrophin (hCG) for women of childbearing potential (WOCBP) (collected only at Screening Visit, and as necessary throughout course of study)

All subjects will have safety laboratory tests at the designated visits outlined in the protocol. These samples will be analyzed at a central laboratory. The Site Investigator (SI) may order additional testing, if needed, to further assess an adverse event (AE), or if there is any suspicion that a subject may be pregnant, throughout the course of the study.

Specific instructions regarding the collection, processing, storage and shipment of these samples will be provided in the Site Manual of Procedures (MOP).

AMX-0035 in ALS Protocol Number: AMX3500


## 8.1.3 Biomarkers and Pharmacokinetic Analysis

Subjects will have blood drawn to assess AMX0035 concentrations for pharmacokinetics (PK) pre-dose at the Baseline Visit and then again at either 1 hour or 4 hours (± 10 minutes) post-dose at the Week 12 and 24 visits. Every attempt should be made to collect samples within the allotted timeframes; however, all samples should be analyzed regardless of actual collection time. The time of administration will be noted. The time of the last meal prior to administration and the time of the drug administration(s) in the previous 24 hours will also be noted.

Additionally, blood will be collected for biomarker analysis, including light and heavy neurofilament testing (NF-L and pNF-H, respectively). Neurofilaments will be used as a mechanistic measure of neuronal death. These proteins are greatly elevated in ALS subjects and promising results from multiple trials suggest this marker may be prognostic of clinical decline. NF-L and pNF-H will be tested over multiple time points with the intention of generating a longitudinal dataset correlating neurofilament levels to observed clinical outcomes. This dataset will help to validate AMX0035 therapeutic mechanism and provide a dataset for the ALS field.

All samples will be labeled with a code. The code will not include any identifiable information. Coded blood samples will be stored at a central laboratory prior to PK and biomarker analysis and other research use.

Specific instructions regarding the collection, processing, storage and shipment of these samples will be provided in the Site Manual of Procedures (MOP).

## 8.1.4 Blood Samples for Future Research Use

Subjects will provide an additional blood sample for storage in a biofluid biorepository at Barrow Neurological Institute. Any research performed on the samples is for research purposes only. These samples will be used for broad future research use in motor neuron diseases. All samples will be labeled with a code. The code will not include any identifiable information. Results of future research will not be provided to the subject or his/her physician.

There is no scheduled date on which the samples will be destroyed. Samples may be stored for research until they are used, damaged, decayed or otherwise unfit for analysis. If a subject no longer wishes to participate in the study and withdraws consent, it will not be possible to destroy samples that may have already been used.

Specific instructions regarding the collection, processing, storage and shipment of these samples will be provided in the Site Manual of Procedures (MOP).

Subjects will have the opportunity to provide an additional optional blood sample for deoxyribonucleic acid (DNA) extraction for genome sequencing at the Baseline Visit. Deidentified blood samples will be sent to the New York Genome Center (NYGC) in New York City, NY.


DNA may be stored, used in genome-wide association studies (GWAS), whole genome sequencing, exome sequencing, or for any other known or as yet undiscovered DNA analysis applicable to understanding or targeting disease, with a particular emphasis on ALS. The information from these genetic studies may be made available to collaborators in academia, not-for-profit settings, or industry for appropriate research. Results of DNA testing from this study will not go into the participant's medical record.

The NYGC will be conducting the sequencing of the coded samples, doing the analysis of the sequencing and sharing the results of such sequencing and analysis with researchers pursuant to this protocol, as well as uploading the data to data repositories such as the National Institutes of Health (NIH) Database of Genotypes and Phenotypes (dbGaP).

## 8.1.5 12-Lead Electrocardiogram (ECG)

A standard 12-lead ECG will be performed. Tracings will be reviewed by a central ECG reader and a copy of the tracings will be kept on site as part of the source documents. The central ECG vendor will provide standard ECG devices for every site and provide training as necessary.

### **8.1.6** Physical Examination

A comprehensive physical examination will be performed and recorded.

## **8.1.7** Neurological Examination

A neurological examination will be performed and recorded. Examination will include assessment of mental status, cranial nerves, motor and sensory function, reflexes, coordination, and stance/gait.

## 8.1.8 Upper Motor Neuron-Burden (UMN-B)

The Penn Upper Motor Neuron-Burden (UMN-B) is the total number of pathological UMN signs on examination including pathologically brisk biceps, supinator, triceps, finger, knee and ankle reflexes, and extensor plantar responses assessed bilaterally and brisk facial and jaw jerks. The scale is a combination of Ashworth, Reflexes, and Pseudobulbar Affect scale (Range score: 0-32).

The UMN also includes scoring of the Center for Neurologic Study-Lability Scale (CNS-LS), a 7-item self-report scale that assesses pseudobulbar affect (PBA) by measuring the perceived frequency of PBA episodes (laughing or crying). Data is generated from the clinical exam and scored from 1-5, the lowest score indicating normal tone and the highest extreme spasticity.

## 8.1.9 Columbia Suicide Severity Rating Scale (C-SSRS)

The US FDA recommends the use of a suicidality assessment instrument that maps to the Columbia Classification Algorithm for Suicide Assessment (C-CASA)<sup>22</sup>. The C-CASA was developed to assist the FDA in coding suicidality data accumulated during the conduct of clinical trials of antidepressant drugs. One such assessment instrument is the Columbia Suicide Severity

AMX-0035 in ALS

Protocol Number: AMX3500


Rating Scale (C-SSRS)<sup>23</sup>. The C-SSRS involves a series of probing questions to inquire about possible suicidal thinking and behavior.

At the Baseline Visit, the C-SSRS Baseline version will be administered. This version is used to assess suicidality over the subject's lifetime.

At all clinic visits after the Baseline Visit, the Since Last Visit version of the C-SSRS will be administered. This version of the scale assesses suicidality since the subject's last visit.

### **8.1.10** Exit Questionnaire

An exit questionnaire will be completed by subjects and Site Investigators at the Final Study Visit (Week 24). This will include questions regarding blindedness and overall experience with the trial.

#### **8.1.11** Adverse Events

Adverse events (AEs) will be documented at each study visit, including the Screening Visit once the informed consent form has been signed by the subject, and at all study visits, including the Final Telephone Call 28 days (+ 5 days) after the last dose of study drug. Information on adverse effects of study drug and on inter-current events will be determined at each visit by direct questioning of the subjects, review of concomitant medications, and vital sign results.

#### 8.2 Outcome Measures

## 8.2.1 ALSFRS-R (Amyotrophic Lateral Sclerosis Functional Rating Scale – Revised)

The ALSFRS-R is a quickly administered (5 minutes) ordinal rating scale (ratings 0-4) used to determine subjects' assessment of their capability and independence in 12 functional activities. All 12 activities are relevant in ALS. Initial validity was established by documenting that in ALS subjects, change in ALSFRS-R scores correlated with change in strength over time, was closely associated with quality of life measures, and predicted survival. The test-retest reliability is greater than 0.88 for all test items. The advantages of the ALSFRS-R are that the categories are relevant to ALS, it is a sensitive and reliable tool for assessing activities of daily living function in those with ALS, and it is quickly administered. With appropriate training the ALSFRS-R can be administered with high inter-rater reliability and test-retest reliability. The ALSFRS-R can be administered by phone with good inter-rater and test-retest reliability. The equivalency of phone versus in-person testing, and the equivalency of study subject versus caregiver responses have also recently been established. The ALSFRS-R will therefore also be given to the study subject over the phone. All ALSFRS-R evaluators must be NEALS certified.

## 8.2.2 Pulmonary Function Testing - Slow Vital Capacity (SVC)

Slow Vital Capacity (SVC): The vital capacity (VC) (percent of predicted normal) will be determined, using the upright slow VC method. The VC can be measured using conventional spirometers that have had a calibration check prior to subject testing. A printout from the

AMX-0035 in ALS Protocol Number: AMX3500

 $Version\ 7.0$ 

spirometer of all VC trials will be retained. All VC evaluators must be NEALS certified. Three VC trials are required for each testing session, however up to 5 trials may be performed if the variability between the highest and second highest VC is 10% or greater for the first 3 trials. Only the 3 best trials are recorded on the CRF. The highest VC recorded is utilized for eligibility.

## **8.2.3** Isometric Strength Testing (ATLIS)

Accurate Testing of Limb Isometric Strength: We are measuring isometric strength using the Accurate Testing of Limb Isometric Strength device (ATLIS) developed by Dr. Patricia Andres of Massachusetts General Hospital. The device was specifically designed to alleviate the reproducibility concerns that exist for prior strength measurements such as hand held dynamometry (HHD). ATLIS does not depend on experimenter strength, and has measurement settings to ensure that subjects are in the same position each time they are tested. All ATLIS evaluators must be trained and certified. ATLIS may detect functional decline before the ALSFRS-R, which may have a ceiling effect, and may be able to detect changes in function with greater sensitivity to ALSFRS-R. The measure does show a small training effect, so we will include measurement at initial screening visit to allow subjects to become acquainted with the device.

## 8.2.4 Neuroimaging MR-PET Sub-Study

A subset of subjects will undergo MR-PET scans at the Baseline Visit and again between the Week 12 and 21 Visits. Prior to the scan, every MR-PET sub-study subject will complete the MR-PET Safety Questionnaire. Scanning procedures and subject instructions will be provided in the Site Manual of Procedures (MOP).

#### 8.2.5 Survival Assessment

Survival endpoint will be considered as mortality, tracheostomy or permanent assisted ventilation.

### 8.2.6 Training and Validation

All evaluators must be NEALS certified to perform the ALSFRS-R, SVC and ATLIS; specific certification requirements are outlined in the study operations manual. Repeat NEALS certification will be required every two years for all NEALS certified outcome measures. It is strongly preferred that a single evaluator performs all measures throughout the study, if possible. NEALS certification is required for all evaluators prior to performing any study tests.

AMX-0035 in ALS Protocol Number: AMX3500


#### SAFETY AND ADVERSE EVENTS

The adverse event (AE) definitions and reporting procedures provided in this protocol comply with all applicable United States Food and Drug Administration (FDA) regulations and International Conference on Harmonization (ICH) guidelines. The Site Investigator will carefully monitor each subject throughout the study for possible adverse events. All AEs will be documented on CRFs designed specifically for this purpose. It is also important to report all AEs, especially those that result in permanent discontinuation of the investigational product being studied, whether serious or non-serious.

#### 9.1 **Definitions of AEs, Suspected Adverse Drug Reactions & SAEs**

## 9.1.1 Adverse Event and Suspected Adverse Drug Reactions

An adverse event (AE) is any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding, for example), symptom, or disease temporally associated with a study, use of a drug product or device whether or not considered related to the drug product or device.

Adverse drug reactions (ADR) are all noxious and unintended responses to a medicinal product related to any dose. The phrase "responses to a medicinal product" means that a causal relationship between a medicinal product and an adverse event is at least a reasonable possibility, i.e., the relationship cannot be ruled out. Therefore, a subset of AEs can be classified as suspected ADRs, if there is a causal relationship to the medicinal product.

Examples of adverse events include: new conditions, worsening of pre-existing conditions, clinically significant abnormal physical examination signs (i.e. skin rash, peripheral edema, etc), or clinically significant abnormal test results (i.e. lab values or vital signs), with the exception of outcome measure results, which are not being recorded as adverse events in this trial (they are being collected, but analyzed separately). Stable chronic conditions (i.e., diabetes, arthritis) that are present prior to the start of the study and do not worsen during the trial are NOT considered adverse events. Chronic conditions that occur more frequently (for intermittent conditions) or with greater severity, would be considered as worsened and therefore would be recorded as adverse events.

Adverse events are generally detected in two ways:

Clinical  $\rightarrow$  symptoms reported by the subject or signs detected on examination.

Ancillary Tests → abnormalities of vital signs, laboratory tests, and other diagnostic procedures (other than the outcome measures, the results of which are not being captured as AEs).


For the purposes of this study, symptoms of progression/worsening of ALS, including 'normal' progression, will be recorded as adverse events.

The following measures of disease progression will not be recorded as adverse events even if they worsen (they are being recorded and analyzed separately): vital capacity results, ALSFRS-R, and ATLIS results.

If discernible at the time of completing the AE log, a specific disease or syndrome rather than individual associated signs and symptoms should be identified by the Site Investigator and recorded on the AE log. However, if an observed or reported sign, symptom, or clinically significant laboratory anomaly is not considered by the Site Investigator to be a component of a specific disease or syndrome, then it should be recorded as a separate AE on the AE log. Clinically significant laboratory abnormalities, such as those that require intervention, are those that are identified as such by the Site Investigator.

Subjects will be monitored for adverse events from the time they sign consent until completion of their participation in the study (defined as death, consent withdrawal, loss to follow up, early study termination for other reasons or following completion of the entire study).

An unexpected adverse event is any adverse event, the specificity or severity of which is not consistent with the current Investigator's Brochure. An unexpected, suspected adverse drug reaction is any unexpected adverse event for which, in the opinion of the Site Investigator or Sponsor (or their designee), there is a reasonable possibility that the investigational product caused the event.

### 9.1.2 Serious Adverse Events

A serious adverse event (SAE) is defined as an adverse event that meets any of the following criteria:

- 1. Results in death.
- 2. Is life threatening: that is, poses an immediate risk of death as the event occurred.
  - a. This serious criterion applies if the study subject, in the view of the Site Investigator or Sponsor, is at immediate risk of death from the AE <u>as it occurs</u>. It does not apply if an AE hypothetically might have caused death if it were more severe.
- 3. Requires in-patient hospitalization or prolongation of existing hospitalization.
  - a. Hospitalization for an elective procedure (including elective PEG tube/g-tube/feeding tube placement) or a routinely scheduled treatment is not an SAE by this criterion because an elective or scheduled "procedure" or a "treatment" is not an untoward medical occurrence.
- 4. Results in persistent or significant disability or incapacity.

AMX-0035 in ALS Protocol Number: AMX3500

 $Version\ 7.0$ 

- a. This serious criterion applies if the "disability" caused by the reported AE results in a substantial disruption of the subject's ability to carry out normal life functions.
- 5. Results in congenital anomaly or birth defect in the offspring of the subject (whether the subject is male or female).
- 6. Necessitates medical or surgical intervention to preclude permanent impairment of a body function or permanent damage to a body structure.
- 7. Important medical events that may not result in death, are not life-threatening, or do not require hospitalization may also be considered SAEs when, based upon appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include blood dyscrasias or convulsions that do not result in in-patient hospitalization, or the development of drug dependency or drug abuse.

An in-patient hospital admission in the absence of a precipitating, treatment-emergent, clinical adverse event may meet criteria for "seriousness" but is not an adverse experience, and will therefore, not be considered an SAE. An example of this would include a social admission (subject admitted for other reasons than medical, e.g., lives far from the hospital, has no place to sleep).

A serious, suspected adverse drug reaction (SUSAR) is an SAE for which, in the opinion of the Site Investigator or Sponsor, there is a reasonable possibility that the investigational product caused the event.

The Site Investigator is responsible for classifying adverse events as serious or non-serious.

## 9.2 Assessment and Recording of Adverse Events

The Site Investigator will carefully monitor each subject throughout the study for possible AEs. All AEs will be documented on source document templates and eCRFs designed specifically for this purpose. All AEs will be collected and reported in the electronic data capture (EDC) system and compiled into reports for periodic reviewing by the Medical Monitor. The Medical Monitor shall promptly review all information relevant to the safety of the investigational product, including all serious adverse events (SAEs). Special attention will be paid to those that result in permanent discontinuation of the investigational product being studied, whether serious or non-serious.

#### 9.2.1 Assessment of Adverse Events

At each visit (including telephone interviews), the subject will be asked if they have had any problems or symptoms since their last visit in order to determine the occurrence of adverse events. If the subject reports an adverse event, the Investigator will probe further to determine:

- 1. Type of event
- 2. Date of onset and resolution (duration)

AMX-0035 in ALS

Protocol Number: AMX3500


- 3. Severity (mild, moderate, severe)
- 4. Seriousness (does the event meet the above definition for an SAE)
- 5. Causality, relation to investigational product and disease
- 6. Action taken regarding investigational product
- 7. Outcome

## 9.2.2 Relatedness of Adverse Event to Investigational Product

The relationship of the AE to the investigational product should be specified by the Site Investigator, using the following definitions:

1. Not Related: Concomitant illness, accident or event with no reasonable

association with treatment.

2. Unlikely: The reaction has little or no temporal sequence from administration

of the investigational product, and/or a more likely alternative

etiology exists.

3. Possibly Related: The reaction follows a reasonably temporal sequence from

administration of the investigational product and follows a known response pattern to the suspected investigational product; the reaction could have been produced by the investigational product or could have been produced by the subject's clinical state or by other modes of therapy administered to the subject. (Suspected

ADR)

4. Probably Related: The reaction follows a reasonably temporal sequence from

administration of investigational product; is confirmed by discontinuation of the investigational product or by re-challenge; and cannot be reasonably explained by the known characteristics

of the subject's clinical state. (Suspected ADR)

5. Definitely Related: The reaction follows a reasonable temporal sequence from

administration of investigational product; that follows a known or expected response pattern to the investigational product; and that is confirmed by improvement on stopping or reducing the dosage of the investigational product, and reappearance of the reaction on

repeated exposure. (Suspected ADR)

AMX-0035 in ALS Protocol Number: AMX3500


## 9.2.3 Adverse Events in Prior Human Experience with Each Individual Component

#### TUDCA

• A small number of subjects (>1%) receiving TUDCA have presented with abdominal discomfort, abdominal pain, diarrhea, nausea, emesis, pruritus, and rash.

#### PB

- O Common adverse events include: menstrual irregularities (23%), decreased appetite (4%), sweat-like body odor (3%), and bad taste (3%)
- Rare effects (<2%) have included Gastrointestinal: abdominal pain, gastritis, nausea and vomiting; constipation, rectal bleeding, peptic ulcer disease, and pancreatitis each occurred in one subject.
  - o Hematologic: aplastic anemia and ecchymoses each occurred in one subject.
  - o Cardiovascular: arrhythmia and edema each occurred in one subject.
  - o Renal: renal tubular acidosis
  - o Psychiatric: depression
  - o Skin: rash
  - o Miscellaneous: headache, syncope, and weight gain
- Hypoalbuminemia, metabolic acidosis, alkalosis, hyperchloremia, hyporhosphatemia, hyporhosphatemia and hypernatremia have been observed.

## 9.2.4 Recording of Adverse Events

All clinical adverse events are recorded in the Adverse Event (AE) Log in the subject's study binder. The site should fill out the AE Log and enter the AE information into the Electronic Data Capture (EDC) system within 48 hours of the site learning of a new AE or receiving an update on an existing AE.

**Please Note:** Serious Adverse Events (SAEs) must be reported to the Medical Monitor and Coordination Center within 24 hours of the site learning of the SAE.

Entries on the AE Log (and into the EDC) will include the following: name and severity of the event, the date of onset, the date of resolution, relationship to investigational product, action taken, and primary outcome of event.

### 9.3 Adverse Events and Serious Adverse Events - Reportable Events

The following are considered reportable events and must be reported to the Medical Monitor and Coordination Center within 24 hours of the site being notified of the event.

o All events that meet the above criteria for Serious Adverse Events (SAEs)

AMX-0035 in ALS

Protocol Number: AMX3500


- Dosage Changes (Dose Management)
  - o Investigational Product Suspension, Reduction or Re-challenge
  - o Investigational Product Discontinuation
- o Key Study Events:
  - Subject Final Disposition
  - o Feeding Tube Placement
  - Permanent Assisted Ventilation (PAV)\*
  - Tracheostomy
  - Mortality
  - o Pregnancy
  - o Diaphragm Pacing System (DPS) device implantation
  - o Emergency or Accidental Unblinding Events
- \* Permanent Assisted Ventilation (PAV) is defined as more than 22 hours daily of non-invasive mechanical ventilation for more than one week (7 days). The date of onset of PAV is the first day of the seven days.


### 10 DATA AND SAFETY MONITORING AND STATISTICAL ANALYSIS PLAN

## 10.1 Data and Safety Monitoring Board

An independent Data and Safety Monitoring Board (DSMB) will be assembled for the trial. The DSMB receives the blinded and unblinded summary reports of the frequency of all clinical adverse events and safety laboratory tests for planned periodic meetings as specified in the DSMB charter. In addition, the DSMB Chair may call ad hoc meetings. Meetings will be held via teleconference. A DSMB Charter will detail the processes of this group.

Summaries of serious adverse events and enrollment will be provided approximately monthly to the DSMB by the Study Biostatisticians. Any possibly, probably or definitely study drug related, serious adverse events (i.e. serious adverse drug reactions, or SUSARs) are considered events of interest and will be reported in real-time (within 1 business day of Coordination Center (CC) awareness) to the DSMB. All adverse events and abnormal laboratory values results will be listed and will be completely identified (using MedDRA adverse reaction codes) by subject and center. The DSMB can ask to receive the SAE reports more frequently. As necessary, the DSMB can review the frequencies of clinical and laboratory abnormalities. Recommendations for modification or termination of the trial based on safety data will be made by the DSMB to the PIs and Steering Committee. The DSMB will review safety data throughout the trial and may stop the trial for safety if they determine that there is a significant difference in the rate of a particular adverse event that would indicate a risk that is greater than the possible benefit of the study drug. A notable increase in the frequency of any adverse event should be examined by the DSMB although it may not lead to a recommendation by the DSMB.

Prior to each DSMB meeting, the CC will provide an update to the DSMB on enrollment, data quality (missing data) and protocol adherence. The CC will be responsible for communication with the DSMB.

Complete information can be found in the Data and Safety Monitoring Board Charter.

#### 10.2 Statistical Considerations

### 10.2.1 Statistical Methods

A challenge in ALS is generating robust data on treatment effects without running prohibitively large studies. Our analysis of the PROACT and ceftriaxone de-identified subject databases suggests that statistical powering can be significantly improved by enrolling subjects who are <1.5 years from symptom onset and have a definite diagnosis of ALS according to El Escorial Criteria . Mixed-effects modeling was used to account for both the variance between subjects and the deviation within subjects from their average rate of decline. We plan to recruit subjects at a rate of at least 10/month to allow for complete enrollment of the study population within 14 months.

AMX-0035 in ALS Protocol Number: AMX3500

Power for safety and tolerability was considered in three ways: incidence of adverse events (AEs), change in ALFSR-R and ATLIS, and change in biomarker such as pNF-H.

With 88 treated subjects, we will have an 80% probability of detecting any adverse event expected to occur in at least 2% of treated subjects. We will have 80% power to detect a 28 percentage point elevation in the rate of any adverse event relative to placebo based on a one-tailed test at alpha = 0.05. We will consider a dose tolerable if the proportion of treatment failures (discontinuation of study drug due to an adverse event) is less than 40% with 80% confidence, one-tailed. With 88 treated subjects this would occur if 30 or fewer subjects on AMX0035 fail to complete the 6-month study. By this criterion, we will have 80% power for declaring AMX0035 tolerable at the tested dose if the true treatment failure rate is 30%.

A shared-baseline, mixed-effects analysis will be used for primary analysis. A covariate of bulbar onset or onset elsewhere and a second covariate of age at enrollment will be included in the analysis. The mixed-effects model accounts for both the variance between subjects and the deviation within subjects from their average rate of decline. We will use the same analysis for clinical outcomes in this trial. We propose to test at an alpha of 0.05.

Further detail on primary analysis and analysis rationale for secondary endpoints will be included in the Statistical Analysis Plan (SAP).

## 10.2.2 Analysis for Safety

The safety data will be summarized by treatment group. Treatment AEs will be coded and graded using MedDRA grading criteria. The treatment groups will be compared with respect to occurrence of each adverse event and incidence of Grade III/IV adverse events. Total number of serious adverse events and abnormal laboratory tests will be compared between groups using Fisher's exact test. Withdrawal, abnormal laboratory tests, vital signs and use of concomitant medications will be assessed to characterize the safety profile of the combination of PB and TUDCA. Compliance data will be determined for each visit and by treatment group. The time to subject refusal will be compared between treatment groups to better determine tolerability. This will be accomplished using a method of survival analysis that allows informative censoring due to death. Descriptive statistics denoting the changes from baseline to the final assessment visit with respect to key laboratory parameters and vital signs will also be provided.

Further detail will be provided in a statistical analysis plan.

AMX-0035 in ALS
Protocol Number: AMX3500


## **10.2.3** Analysis for Efficacy

Modified intention-to-treat analysis will be performed, including all randomized subjects receiving at least one dose of the study medication and having at least one primary efficacy assessment after randomization. Slope will be imputed from available data and time points. Homogeneity of clinical characteristics and efficacy variables at baseline between the two randomization groups (between-group baseline differences) will be assessed by analysis of variance for continuous variables and by a chi-squared test for discrete variables. All efficacy endpoints will compared between the two randomization groups at study end (between-group differences at study end) by means of analysis of covariance for continuous variables, adjusting for baseline value and for center effect, and by a chi-squared test for discrete variables. Survival time will compared between treatments by a Kaplan–Meier survival analysis.

The primary analysis strategy will use a shared-baseline, mixed-effects model of ALSFRS-R progression rate. The mixed-effects model accounts for both the variance between subjects and the deviation within subjects from their average rate of decline. We will use the same analysis for clinical outcomes in this trial. We propose to test at an alpha of 0.05. We are targeting an effect size (slowing of ALSFRS-R slope) greater than 30% based on the trial by Elia et al<sup>17</sup>. In the Phase I/II trial of TUDCA that analyzed a total of 29 subjects, the ALSFRS-R score declined 32.5% more slowly in the TUDCA group: the slopes of the two regression lines were significantly different (-0.262/week for the TUDCA group, -0.388/week for the placebo group; P < 0.01).

# 10.2.4 Analysis Populations

The modified intent to treat (ITT) population will include all study subjects who are randomized and receive at least one dose of study drug. The ITT population will be considered for primary analyses. For ITT analyses, subjects will be grouped based on randomized treatment, regardless of treatment actually received.

## 10.3 Missing Data

The trial will be modified intent to treat (ITT). Every effort will be made to obtain follow-up information for all subjects whether or not they continue on treatment.


## 11 DATA COLLECTION, MANAGEMENT AND MONITORING

# 11.1 Role of Data Management

Data Management (DM) is the development, execution and supervision of plans, policies, programs, and practices that control, protect, deliver, and enhance the value of data and information assets.

All data will be managed in compliance with applicable Sponsor (or their designee) policies and regulatory requirements. Site personnel will collect, transcribe, correct, and transmit the data onto source documents, Case Report Forms (CRFs), and other forms used to report, track and record clinical research data. Clinical sites will be monitored to ensure compliance with data management requirements and Good Clinical Practices. DM is responsible for developing, testing, and managing clinical data management activities.

# 11.1.1 Data Entry and Checks

The site personnel are encouraged to enter information into the Electronic Data Capture (EDC) System within 5 days of a visit. Please Note: Serious Adverse Events (SAEs) must be reported to the Coordination Center within 24 hours of the site learning of the SAE. Data collection is the responsibility of the staff at the site under the supervision of the Site Investigator (SI). During the study, the Site Investigator must maintain complete and accurate documentation for the study.

The EDC includes password protection. An edit checking and data clarification process will be put in place to ensure accuracy and completeness of the database. Logic and range checks as well as more sophisticated rules will be built into the EDC to provide immediate error checking of the data entered. The system has the capability to automatically create electronic queries for forms that contain data that are out of range, out of window, missing or not calculated correctly. The sites will only have access to the queries concerning their subjects.

## 11.1.2 Data Lock Process

The application will have the ability to lock the database to prevent any modification of data once the study is closed. Once this option is activated, every user will have Read-Only access to the data. The database can only be locked after each Site Investigator (SI) has signed off on their subjects and all queries have been resolved.

## 11.1.3 Quality Assurance

Protocol procedures are reviewed with the Site Investigator (SI) and associated personnel prior to the study to ensure the accuracy and reliability of data. Each SI must adhere to the protocol detailed in this document and agree that any changes to the protocol must be approved by the Coordination Center prior to seeking approval from the central IRB. Each Site Investigator will be responsible for enrolling only those study subjects who have met protocol eligibility criteria.

AMX-0035 in ALS Protocol Number: AMX3500


# 11.2 Clinical Monitoring

Study Monitors will visit each study site to review source documentation materials, informed consent forms, and confirm entered data and that data queries have been accurately completed, and again at a study close-out visit. Study Monitors will also verify that SAEs and protocol deviations have been reported appropriately, as required. The Study Monitors will also review clinical facilities, resources and procedures for evaluating study subjects and study drug dispensing. Subsequently, the Study Monitors will provide monitoring reports to the Project Manager and, if requested, will provide reports of protocol compliance to the Study Principal Investigator and the Steering Committee. Completed informed consent forms from each subject must be available in the subject's file and verified for proper documentation. A document outlining the monitoring plan is provided to each Study Monitor.

## 11.3 Data Handling and Record Keeping

The Site Investigator (SI) is responsible to ensure the accuracy, completeness, legibility, and timeliness of the data reported. All source documents should be completed in a neat, legible manner to ensure accurate interpretation of data. Dark ink is required to ensure clarity of reproduced copies. When making changes or corrections, cross out the original entry with a single line, and initial and date the change. Do not erase, overwrite, or use correction fluid or tape on the original.

Source document templates (SDTs) will be provided for use and maintained for recording data for each subject enrolled in the study. Data reported in the eCRF derived from source documents should be consistent with the source documents and discrepancies should be explained. The Coordination Center will provide guidance to SIs on making corrections to the source documents and eCRFs.

### 11.3.1 Confidentiality

Study subject medical information obtained by this study is confidential, and disclosure to third parties other than those noted below is prohibited. Upon the subject's permission, medical information may be given to his or her personal physician or other appropriate medical personnel responsible for his or her welfare. All local and federal guidelines and regulations regarding maintaining study subject confidentiality of data will be adhered to.

Data generated by this study must be available for inspection by representatives of the US FDA, the Office for Human Research Protections (OHRP), the Sponsor, all pertinent national and local health and regulatory authorities, the Coordination Center or their representative, Study Monitoring personnel, and the central IRB.

## 11.3.2 Study Discontinuation

The study can be terminated at any time by the Sponsor, DSMB, or FDA. Reasons for terminating the study may include the following:

• The incidence or severity of AEs in this or other studies indicates a potential health hazard to study subjects.

AMX-0035 in ALS

Protocol Number: AMX3500


- Study subject enrollment is unsatisfactory.
- Data recording is inaccurate or incomplete.
- Sponsor withdraws funding.

### 11.3.3 Retention of Records

US FDA regulations (21 CFR 312.62[c]) require that records and documents pertaining to the conduct of this study and the distribution of investigational drug, including CRFs (if applicable), consent forms, laboratory test results, and medical inventory records, must be retained by the Site Investigator (SI) for two years after marketing application approval. If no application is filed, these records must be kept for two years after the investigation is discontinued and the US FDA and the applicable national and local health authorities are notified. The Coordination Center or their representative will notify the Site Investigators of these events. The Site Investigators should retain all study documents and records until they are notified in writing by the Sponsor or their representative.

## 11.3.4 Publications

The Study Principal Investigator, , along with the Sponsor, Amylyx Pharmaceuticals, Inc., will be responsible for publications of results from this trial. Their responsibilities will include the following:

- Analyze and interpret data gathered in this study, and write publications from these data.
- Submit manuscripts to selected journals and address peer reviewers' comments.
- Submit abstracts to selected meetings and present data at the meetings.
- Determine authorship on the basis of the Uniform Requirements for Manuscripts.


## 12 LITERATURE REFERENCES

- 1. Manfredi, G and Kawamata, H Mitochondria and endoplasmic reticulum crosstalk in amyotrophic lateral sclerosis. Neurobiology of Disease. 2015.
- 2. Zhou, W et al. Phenylbutyrate up-regulates the DJ-1 protein and protects neurons in cell culture and in animal models of Parkinson disease. J Biol Chem. 2011.
- 3. Suaud, L et Al. ERp29 Regulates F508 and Wild-type Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) Trafficking to the Plasma Membrane in Cystic Fibrosis (CF) and Non-CF Epithelial Cells. JBC. 2011
- 4. Ryu, H et al. Sodium phenylbutyrate prolongs survival and regulates expression of antiapoptotic genes in transgenic amyotrophic lateral sclerosis mice. J Neurochem. 2005.
- 5. Gardian G, Browne SE, Choi DK, Klivenyi P, Gregorio J, Kubilus JK, Ryu H, Langley B, Ratan RR, Ferrante RJ, et al. Neuroprotective effects of phenylbutyrate in the N171-82Q transgenic mouse model of Huntington's disease. J Biol Chem. 2005
- 6. Ricobaraza A, Cuadrado-Tejedor M, Pérez-Mediavilla A, Frechilla D, Del Río J, García-Osta A. Phenylbutyrate ameliorates cognitive deficit and reduces tau pathology in an Alzheimer's disease mouse model. Neuropsychopharmacology. 2009
- 7. Roy, A, et al. Sodium Phenylbutyrate Controls Neuroinflammatory and Antioxidant Activities and Protects Dopaminergic Neurons in Mouse Models of Parkinson's Disease. PLoS ONE. 2012.
- 8. Rodrigues, CM. et al. Tauroursodeoxycholic acid prevents Bax-induced membrane perturbation and cytochrome C release in isolated mitochondria. Biochemistry. 2003.
- 9. Zhang et al. Aggregation-prone c9FTD/ALS poly(GA) RAN-translated proteins cause neurotoxicity by inducing ER stress. Acta Neuropath 2014
- 10. Rodrigues et al. Tauroursodeoxycholic acid reduces apoptosis and protects against neurological injury after acute hemorrhagic stroke in rats. PNAS. 2003.
- 11. Castro-Caldas et al. Tauroursodeoxycholic acid prevents MPTP-induced dopaminergic cell death in a mouse model of Parkinson's disease. J. Mol. Neurobiol. 2012
- 12. Lewis CA, Manning J, Rossi F, Krieger C. The Neuroinflammatory Response in ALS: The Roles of Microglia and T Cells. Neurol Res Int 2012;2012:803701.
- 13. Huang Y, Henry CJ, Dantzer R, Johnson RW, Godbout JP. Exaggerated sickness behavior and brain proinflammatory cytokine expression in aged mice in response to intracerebroventricular lipopolysaccharide. Neurobiol Aging 2008;29:1744-53.
- 14. Berger A. Th1 and Th2 responses: what are they? BMJ 2000;321:424.
- 15. Cudkowicz, ME et al. Phase 2 study of sodium phenylbutyrate in ALS. Amyotrophic Lateral Sclerosis. 2009.
- 16. Hogarth, P. et al. Sodium Phenylbutyrate in Huntington's Disease: A Dose-Finding Study. Movement Disorders. 2007.
- 17. Elia, AE et al. Tauroursodeoxycholic acid in the treatment of subjects with amyotrophic lateral sclerosis. Eur J. Neurol. 2015.

AMX-0035 in ALS

Protocol Number: AMX3500


- 18. Min, JH et al. Oral Solubilized Ursodeoxycholic Acid Therapy in Amyotrophic Lateral Sclerosis: A Randomized Cross-Over Trial. J. Korean Medical Science. 2012.
- 19. Buphenyl Package Insert
- 20. Gilbert, J. et al. A phase I dose escalation and bioavailability study of oral sodium phenylbutyrate in patients with refractory solid tumor malignancies. Clin Cancer Res. 2001.
  - Gore, SD et al. Impact of the putative differentiating agent sodium phenylbutyrate on myelodysplastic syndromes and acute myeloid leukemia. Clin Cancer Res. 2001.
- 21. Zurcher et al. Increased in vivo glial activation in subjects with amyotrophic lateral sclerosis: Assessed with [11C]-PBR28. Neuroimage Clin. 2015.
- 22. Posner K, (et.al), Columbia Classification Algorithm of Suicide Assessment (C-CASA): Classification of Suicidal Events in the FDA's Pediatric Suicidal Risk Analysis of Antidepressants, Am J Psychiatry, 2007, 164:1035-1043.
- 23. September 2010 US FDA Draft Guidance for Industry Suicidality: Prospective Assessment of Occurrence in Clinical Trials

#### 13 APPENDICES

# 13.1 APPENDIX I: EL ESCORIAL WORLD FEDERATION OF NEUROLOGY CRITERIA FOR THE DIAGNOSIS OF ALS

Information obtained from the web site: www.wfnals.org.

The diagnosis of Amyotrophic Lateral Sclerosis [ALS] requires:

## A - The presence of:

- (A:1) evidence of lower motor neuron (LMN) degeneration by clinical, electrophysiology or neuropathologic examination,
- (A:2) evidence of upper motor neuron (UMN) degeneration by clinical examination, and
- (A:3) progressive spread of symptoms or signs within a region or to other regions, as determined by history or examination, together with

## B - The absence of:

- (B:1) electrophysiological and pathological evidence of other disease processes that might explain the signs of LMN and/or UMN degeneration, and
- (B:2) neuroimaging evidence of other disease processes that might explain the observed clinical and electrophysiological signs.

## CLINICAL STUDIES IN THE DIAGNOSIS OF ALS

A careful history, physical and neurological examination must search for clinical evidence of UMN and LMN signs in four regions [brainstem, cervical, thoracic, or lumbosacral spinal cord] (see Table 1) of the central nervous system [CNS]. Ancillary tests should be reasonably applied, as clinically indicated, to exclude other disease processes. These should include electrodiagnostic, neurophysiological, neuroimaging and clinical laboratory studies. Clinical evidence of LMN and UMN degeneration is required for the diagnosis of ALS. The clinical diagnosis of ALS, without pathological confirmation, may be categorized into various levels of certainty by clinical assessment alone depending on the presence of UMN and LMN signs together in the same topographical anatomic region in either the brainstem [bulbar cranial motor neurons], cervical, thoracic, or lumbosacral spinal cord [anterior horn motor neurons]. The terms Clinical Definite ALS and Clinically Probable ALS are used to describe these categories of clinical diagnostic certainty on clinical criteria alone:

- A. Clinically Definite ALS is defined on clinical evidence alone by the presence of UMN, as well as LMN signs, in three regions.
- B. Clinically Probable ALS is defined on clinical evidence alone by UMN and LMN signs in at least two regions with some UMN signs necessarily rostral to (above) the LMN signs.

AMX-0035 in ALS

Protocol Number: AMX3500


C. Clinically Probable ALS - Laboratory-supported is defined when clinical signs of UMN and LMN dysfunction are in only one region, or when UMN signs alone are present in one region, and LMN signs defined by EMG criteria are present in at least two limbs, with proper application of neuroimaging and clinical laboratory protocols to exclude other causes.

D. Clinically Possible ALS is defined when clinical signs of UMN and LMN dysfunction are found together in only one region or UMN signs are found alone in two or more regions; or LMN signs are found rostral to UMN signs and the diagnosis of Clinically Probable - Laboratory-supported ALS cannot be proven by evidence on clinical grounds in conjunction with electrodiagnostic, neurophysiologic, neuroimaging or clinical laboratory studies. Other diagnoses must have been excluded to accept a diagnosis of Clinically Possible ALS.

Table 1

| | Brainstem | Cervical | Thoracic | Lumbosacral |
|---|---|---|---|---|
| Lower motor<br>neuron signs<br>weakness,<br>atrophy,<br>fasciculations | jaw, face,<br>palate,<br>tongue, larynx | neck, arm, hand, diaphragm | back,<br>abdomen | back, abdomen,<br>leg, foot |
| Upper motor<br>neuron signs<br>pathologic spread<br>of reflexes, clonus,<br>etc. | clonic jaw gag reflex exaggerated snout reflex pseudobulbar features forced yawning pathologic DTRs spastic tone | clonic DTRs Hoffman reflex pathologic DTRs spastic tone preserved reflex in weak wasted limb | loss of<br>superficial<br>abdominal<br>reflexes<br>pathologic<br>DTRs<br>spastic tone | clonic DTRs - extensor plantar response pathologic DTRs spastic tone preserved reflex in weak wasted limb |

AMX-0035 in ALS Protocol Number: AMX3500


# 13.2 APPENDIX II: ALS FUNCTIONAL RATING SCALE – REVISED (ALSFRS-R) ALSFRS-R

| QUESTIONS: | <b>SCORE:</b> |
|---|---|
| 1. Speech | |
| 4 = Normal speech processes | |
| 3 = Detectable speech disturbances | |
| 2 = Intelligible with repeating | |
| 1 = Speech combined with nonvocal communication | |
| 0 = Loss of useful speech | |
| 2. Salivation | |
| 4 = Normal | |
| 3 = Slight but definite excess of saliva in mouth; may have nighttime | drooling |
| 2 = Moderately excessive saliva; may have minimal drooling | |
| 1 = Marked excess of saliva with some drooling | |
| 0 = Marked drooling; requires constant tissue or handkerchief | |
| 2.6.11 | |
| 3. Swallowing | |
| 4 = Normal eating habits | |
| 3 = Early eating problems – occasional choking | |
| 2 = Dietary consistency changes<br>1 = Needs supplemental tube feeding | |
| 0 = NPO (exclusively parenteral or enteral feeding) | |
| 0 – IN O (exclusively parenteral of enteral recuing) | |
| 4. Handwriting | |
| 4 = Normal | |
| 3 = Slow or sloppy; all words are legible | |
| 2 = Not all words are legible | |
| 1 = No words are legible but can still grip a pen | |
| 0 = Unable to grip pen | |
| | ` |
| 5a. Cutting Food and Handling Utensils (subjects without gastrostomy | y) |
| 4 = Normal | |
| 3 = Somewhat slow and clumsy, but no help needed | 1 |
| 2 = Can cut most foods, although clumsy and slow; some help needed | L |
| 1 = Food must be cut by someone, but can still feed slowly | |

AMX-0035 in ALS

Protocol Number: AMX3500

0 =Needs to be fed


| 5b. Cutting Food and Handling Utensils (alternate scale for subjects with gastrostomy) |
|---|
| 4 = Normal |
| 3 = Clumsy, but able to perform all manipulations independently 2 = Some help needed with closures and fasteners 1 = Provides minimal assistance to caregivers 0 = Unable to perform any aspect of task |
| 6. Dressing and Hygiene 4 = Normal function 3 = Independent, can complete self-care with effort or decreased efficiency 2 = Intermittent assistance or substitute methods 1 = Needs attendant for self-care 0 = Total dependence |
| 7. Turning in Bed and Adjusting Bed Clothes 4 = Normal function 3 = Somewhat slow and clumsy, but no help needed 2 = Can turn alone, or adjust sheets, but with great difficulty 1 = Can initiate, but not turn or adjust sheets alone 0 = Helpless |
| 8. Walking 4 = Normal 3 = Early ambulation difficulties 2 = Walks with assistance 1 = Nonambulatory functional movement only 0 = No purposeful leg movement |
| <ul> <li>9. Climbing Stairs</li> <li>4 = Normal</li> <li>3 = Slow</li> <li>2 = Mild unsteadiness or fatigue</li> <li>1 = Needs assistance</li> </ul> |

AMX-0035 in ALS

0 = Cannot do

Protocol Number: AMX3500


| R-1. Dyspnea | |
|---|---|
| 4 = None | |
| 3 = Occurs when walking | |
| 2 = Occurs with one or more of the following: eating, bathing, dressing | |
| 1 = Occurs at rest, difficulty breathing when either sitting or lying | |
| 0 = Significant difficulty, considering using mechanical respiratory support | |
| R-2 Orthopnea | |
| 4 = None | |
| 3 = Some difficulty sleeping at night due to shortness of breath, does not routinely use | more than |
| two pillows | |
| 2 = Needs extra pillow in order to sleep (more than two) | |
| 1 = Can only sleep sitting up | |
| 0 = Unable to sleep without mechanical assistance | |
| R-3 Respiratory Insufficiency | |
| 4 = None | |
| 3 = Intermittent use of BiPAP | |
| 2 = Continuous use of BiPAP during the night | |
| 1 = Continuous use of BiPAP during the night and day | |
| 0 = Invasive mechanical ventilation by intubation or tracheostomy | |
| Evaluator's Initials: | |

AMX-0035 in ALS Protocol Number: AMX3500


# 13.3 APPENDIX III: COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS) BASELINE VERSION

Information obtained from: http://www.cssrs.columbia.edu/

| SUICIDAL IDEATION | |
|---|---|
| Ask questions 1 and 2. If both are negative, proceed to "Suicidal Behavior" section. If the answer to question 2 is "yes", ask questions 3, 4 and 5. If the answer to question 1 and/or 2 is "yes", complete "Intensity of Ideation" section below. | Lifetime:<br>Time<br>He/She<br>Felt Most<br>Suicidal |
| 1. Wish to be Dead | Yes No |
| Subject endorses thoughts about a wish to be dead or not alive anymore, or wish to fall asleep and not wake up. | |
| Have you wished you were dead or wished you could go to sleep and not wake up? If yes, describe: | |
| 2. Non-Specific Active Suicidal Thoughts | Yes No |
| General, non-specific thoughts of wanting to end one's life/commit suicide (e.g., "I've thought about killing myself") without thoughts of ways to kill oneself/associated methods, intent, or plan. Have you actually had any thoughts of killing yourself? | |
| If yes, describe: | |
| 3. Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act | Yes No |
| Subject endorses thoughts of suicide and has thought of at least one method during the assessment period. This is different than a specific plan with time, place or method details worked out (e.g., thought of method to | |
| kill self but not a specific plan). Includes person who would say, "I thought about taking an overdose but I never made a specific plan as to when, where or how I would actually do itand I would never go through with | |
| it." | |
| Have you been thinking about how you might do this? If yes, describe: | |
| 4. Active Suicidal Ideation with Some Intent to Act, without Specific Plan | Yes No |
| Active suicidal thoughts of killing oneself and subject reports having some intent to act on such thoughts, as | Yes No |
| Active suicidal thoughts of killing oneself and subject reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them." | |
| Active suicidal thoughts of killing oneself and subject reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them." Have you had these thoughts and had some intention of acting on them? | |
| Active suicidal thoughts of killing oneself and subject reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them." Have you had these thoughts and had some intention of acting on them? If yes, describe: 5. Active Suicidal Ideation with Specific Plan and Intent Thoughts of killing oneself with details of plan fully or partially worked out and subject has some intent to carry | |
| Active suicidal thoughts of killing oneself and subject reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them." Have you had these thoughts and had some intention of acting on them? If yes, describe: 5. Active Suicidal Ideation with Specific Plan and Intent Thoughts of killing oneself with details of plan fully or partially worked out and subject has some intent to carry it out. Have you started to work out or worked out the details of how to kill yourself? Do you intend to carry | ☐ ☐ Yes No |
| Active suicidal thoughts of killing oneself and subject reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them." Have you had these thoughts and had some intention of acting on them? If yes, describe: 5. Active Suicidal Ideation with Specific Plan and Intent Thoughts of killing oneself with details of plan fully or partially worked out and subject has some intent to carry it out. | ☐ ☐ Yes No |
| Active suicidal thoughts of killing oneself and subject reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them." Have you had these thoughts and had some intention of acting on them? If yes, describe: 5. Active Suicidal Ideation with Specific Plan and Intent Thoughts of killing oneself with details of plan fully or partially worked out and subject has some intent to carry it out. Have you started to work out or worked out the details of how to kill yourself? Do you intend to carry out this plan? If yes, describe: INTENSITY OF IDEATION | ☐ ☐ Yes No |
| Active suicidal thoughts of killing oneself and subject reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them." Have you had these thoughts and had some intention of acting on them? If yes, describe: 5. Active Suicidal Ideation with Specific Plan and Intent Thoughts of killing oneself with details of plan fully or partially worked out and subject has some intent to carry it out. Have you started to work out or worked out the details of how to kill yourself? Do you intend to carry out this plan? If yes, describe: INTENSITY OF IDEATION The following features should be rated with respect to the most severe type of ideation (i.e., 1-5) | Yes No |
| Active suicidal thoughts of killing oneself and subject reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them." Have you had these thoughts and had some intention of acting on them? If yes, describe: 5. Active Suicidal Ideation with Specific Plan and Intent Thoughts of killing oneself with details of plan fully or partially worked out and subject has some intent to carry it out. Have you started to work out or worked out the details of how to kill yourself? Do you intend to carry out this plan? If yes, describe: INTENSITY OF IDEATION | Yes No |
| Active suicidal thoughts of killing oneself and subject reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them." Have you had these thoughts and had some intention of acting on them? If yes, describe: 5. Active Suicidal Ideation with Specific Plan and Intent Thoughts of killing oneself with details of plan fully or partially worked out and subject has some intent to carry it out. Have you started to work out or worked out the details of how to kill yourself? Do you intend to carry out this plan? If yes, describe: INTENSITY OF IDEATION The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. | Yes No |
| Active suicidal thoughts of killing oneself and subject reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them." Have you had these thoughts and had some intention of acting on them? If yes, describe: 5. Active Suicidal Ideation with Specific Plan and Intent Thoughts of killing oneself with details of plan fully or partially worked out and subject has some intent to carry it out. Have you started to work out or worked out the details of how to kill yourself? Do you intend to carry out this plan? If yes, describe: INTENSITY OF IDEATION The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she | Yes No |
| Active suicidal thoughts of killing oneself and subject reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them." Have you had these thoughts and had some intention of acting on them? If yes, describe: 5. Active Suicidal Ideation with Specific Plan and Intent Thoughts of killing oneself with details of plan fully or partially worked out and subject has some intent to carry it out. Have you started to work out or worked out the details of how to kill yourself? Do you intend to carry out this plan? If yes, describe: INTENSITY OF IDEATION The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Most Severe Ideation: Type # (1-5) Description of Ideation Frequency | Yes No |
| Active suicidal thoughts of killing oneself and subject reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them." Have you had these thoughts and had some intention of acting on them? If yes, describe: 5. Active Suicidal Ideation with Specific Plan and Intent Thoughts of killing oneself with details of plan fully or partially worked out and subject has some intent to carry it out. Have you started to work out or worked out the details of how to kill yourself? Do you intend to carry out this plan? If yes, describe: INTENSITY OF IDEATION The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Most Severe Ideation: Type # (1-5) Description of Ideation | Yes No |

AMX-0035 in ALS Protocol Number: AMX3500


| Duration |
|---|
| When you have the thoughts, how long do they last? |
| (1) Fleeting - few seconds or minutes (4) 4-8 hours/most of day |
| (2) Less than 1 hour/some of the time (5) More than 8 hours/persistent or continuous |
| (3) 1-4 hours/a lot of time |
| Controllability |
| Could/can you stop thinking about killing yourself or wanting to die if you want to? |
| (1) Easily able to control thoughts (4) Can control thoughts with a lot of difficulty |
| (2) Can control thoughts with little difficulty (5) Unable to control thoughts |
| (3) Can control thoughts with some difficulty (0) Does not attempt to control thoughts |
| Deterrents |
| Are there things - anyone or anything (e.g., family, religion, pain of death) - that |
| stopped you from wanting to die or acting on thoughts of committing suicide? |
| (1) Deterrents definitely stopped you from attempting suicide (4) Deterrents most likely did not stop you |
| (2) Deterrents probably stopped you (5) Deterrents definitely did not stop you |
| (3) Uncertain that deterrents stopped you (0) Does not apply |
| Reasons for Ideation |
| What sort of reasons did you have for thinking about wanting to die or killing |
| yourself? Was it to end the pain or stop the way you were feeling (in other words you |
| couldn't go on living with this pain or how you were feeling) or was it to get attention, |
| revenge or a reaction from others? Or both? |
| (1) Completely to get attention, revenge or a reaction from others (4) Mostly to end or stop the pain (you |
| couldn't go on |
| (2) Mostly to get attention, revenge or a reaction from others living with the pain or how you were feeling) |
| (3) Equally to get attention, revenge or a reaction from others (5) Completely to end or stop the pain (you |
| couldn't go on |
| and to end/stop the pain. living with the pain or how you were feeling) |
| (0) Does not apply |

| SUICIDAL BEHAVIOR | Lifetime |
|---|---|
| (Check all that apply, so long as these are separate events; must ask about all types) | |
| Actual Attempt: | Yes No |
| A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in | пп |
| part thought of as method to kill oneself. Intent does not have to be 100%. If there is <b>any</b> intent/desire to die | |
| associated with the act, then it can be considered an actual suicide attempt. <i>There does not have to be</i> | Total # of |
| any injury or harm, just the potential for injury or harm. If person pulls trigger while gun is in mouth but | Attempts |
| gun is broken so no injury results, this is considered an attempt. | |
| Inferring Intent: Even if an individual denies intent/wish to die, it may be inferred clinically from the behavior or | |
| circumstances. For example, a highly lethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping from window of a high floor/story). Also, if someone denies | Yes No |
| intent to die, but they thought that what they did could be lethal, intent may be inferred. | |
| Have you made a suicide attempt? | |
| Have you done anything to harm yourself? | |
| Have you done anything dangerous where you could have died? | |
| What did you do? | |
| Did you as a way to end your life? | |
| Did you want to die (even a little) when you? | |
| Were you trying to end your life when you? | |
| Or did you think it was possible you could have died from? | |
| Or did you do it purely for other reasons / without ANY intention of killing yourself (like | |
| to relieve stress, feel better, get sympathy, or get something else to happen)? (Self- | |
| Injurious Behavior without suicidal intent) | |
| If yes, describe: | |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? | |

AMX-0035 in ALS

Protocol Number: AMX3500


| Interrupted Attempt: | | | Yes No |
|---|---|---|---|
| When the person is interrupted (by an outside circumstance) from starting the potent not for that, actual attempt would have occurred). | ially self-injuri | ous act (if | |
| Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt. Shooting: Person has gun pointed toward self, gun is taken away by someone else, or is somehow prevented from pulling trigger. Once they pull the trigger, even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken down from ledge. Hanging: Person has noose around neck but has not yet started to hang - is stopped from doing so. | | aken away<br>the gun<br>dge. | Total # of interrupted |
| Hanging: Person has noose around neck but has not yet started to hang - is stopped<br>Has there been a time when you started to do something to end you | | | |
| or something stopped you before you actually did anything? | ur me but | Someone | |
| If yes, describe: | | | |
| Aborted Attempt: | | | Yes No |
| When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of being stopped by something else. | | | |
| Has there been a time when you started to do something to try to | end your lif | e but | Total # of<br>aborted |
| you stopped yourself before you actually did anything? | | | |
| If yes, describe: | | | |
| Preparatory Acts or Behavior: | | | Yes No |
| Acts or preparation towards imminently making a suicide attempt. This can include a verbalization or thought, such as assembling a specific method (e.g., buying pills, pu preparing for one's death by suicide (e.g., giving things away, writing a suicide note). | rchasing a gu | d a<br>n) or | |
| Have you taken any steps towards making a suicide attempt or pre | | kill | |
| yourself (such as collecting pills, getting a gun, giving valuables a | way or wri | ting a | |
| suicide note)? | | | |
| If yes, describe: Suicidal Behavior: | | | Yes No |
| Suicidal behavior was present during the assessment period? | | | |
| Answer for Actual Attempts Only | Most | Most | Initial/First |
| / | Recent | Lethal | Attempt<br>Date: |
| | Attempt<br>Date: | Attempt<br>Date: | Date. |
| Actual Lethality/Medical Damage: | Enter | Enter | Enter Code |
| No physical damage or very minor physical damage (e.g., surface scratches). Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). | Code<br>——— | Code<br>——— | |
| Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major | | | |
| vessel). 3. Moderately severe physical damage; <i>medical</i> hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less | | | |
| than 20% of body; extensive blood loss but can recover; major fractures). | | | |
| 4. Severe physical damage; <i>medical</i> hospitalization with intensive care required | | | |
| (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). | | | |
| 5. Death | | | |
| Potential Lethality: Only Answer if Actual Lethality=0 | Enter | Enter | Enter Code |
| Likely lethality of actual attempt if no medical damage (the following examples, | Code | Code | |
| while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; | | | |
| laying on train tracks with oncoming train but pulled away before run over). | | | |
| 0 = Behavior not likely to result in injury 1 = Behavior likely to result in injury but not likely to cause death | | | |
| 2 = Behavior likely to result in death despite available medical care | | | |


# 13.4 APPENDIX IV: COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS) SINCE LAST VISIT VERSION

Information obtained from: http://www.cssrs.columbia.edu/

| SUICIDAL IDEATION | |
|---|---|
| Ask questions 1 and 2. If both are negative, proceed to "Suicidal Behavior" section. If the | Since |
| answer to question 2 is "yes", ask questions 3, 4 and 5. If the answer to question 1 and/or 2 is | Last |
| "yes", complete "Intensity of Ideation" section below. | Visit |
| 1. Wish to be Dead | Yes No |
| Subject endorses thoughts about a wish to be dead or not alive anymore, or wish to fall asleep and not wake up. | |
| Have you wished you were dead or wished you could go to sleep and not wake up? | |
| If yes, describe: | |
| 2. Non-Specific Active Suicidal Thoughts | Yes No |
| General, non-specific thoughts of wanting to end one's life/commit suicide (e.g., "I've thought about killing myself") | |
| without thoughts of ways to kill oneself/associated methods, intent, or plan during the assessment period. | |
| Have you actually had any thoughts of killing yourself? If yes, describe: | |
| 3. Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act | Yes No |
| Subject endorses thoughts of suicide and has thought of at least one method during the assessment period. This is different than a specific plan with time, place or method details worked out (e.g., thought of method to kill self but not a | |
| specific plan). Includes person who would say, "I thought about taking an overdose but I never made a specific plan as | |
| to when, where or how I would actually do itand I would never go through with it." | |
| Have you been thinking about how you might do this? | |
| If yes, describe: | Vac Na |
| 4. Active Suicidal Ideation with Some Intent to Act, without Specific Plan | Yes No |
| Active suicidal thoughts of killing oneself and subject reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them." | |
| Have you had these thoughts and had some intention of acting on them? | |
| If yes, describe: | |
| 5. Active Suicidal Ideation with Specific Plan and Intent | Yes No |
| Thoughts of killing oneself with details of plan fully or partially worked out and subject has some intent to carry it out. | |
| Have you started to work out or worked out the details of how to kill yourself? Do you intend to carry out this | |
| plan? | |
| If yes, describe: | |
| INTENSITY OF IDEATION | , |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from | Most |
| above, with 1 being the least severe and 5 being the most severe). | Severe |
| Most Severe Ideation: | |
| Type # (1-5) Description of Ideation | |
| Frequency | |
| How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day | |
| Duration | |
| When you have the thoughts, how long do they last? | |
| (1) Fleeting - few seconds or minutes (4) 4-8 hours/most of day | |
| (2) Less than 1 hour/some of the time (5) More than 8 hours/persistent or continuous | |
| (3) 1-4 hours/a lot of time | |
| Controllability | |
| Could/can you stop thinking about killing yourself or wanting to die if you want to? | |
| (1) Easily able to control thoughts (4) Can control thoughts with a lot of difficulty | |
| (2) Can control thoughts with little difficulty (5) Unable to control thoughts (3) Can control thoughts with some difficulty (0) Does not attempt to control thoughts | |

AMX-0035 in ALS

Protocol Number: AMX3500


| Deterrents |
|---|
| Are there things - anyone or anything (e.g., family, religion, pain of death) - that stopped you |
| from wanting to die or acting on thoughts of committing suicide? |
| (1) Deterrents definitely stopped you from attempting suicide (4) Deterrents most likely did not stop you |
| (2) Deterrents probably stopped you (5) Deterrents definitely did not stop you |
| (3) Uncertain that deterrents stopped you (0) Does not apply |
| Reasons for Ideation |
| What sort of reasons did you have for thinking about wanting to die or killing yourself? Was |
| it to end the pain or stop the way you were feeling (in other words you couldn't go on living |
| with this pain or how you were feeling) or was it to get attention, revenge or a reaction from |
| others? Or both? |
| (1) Completely to get attention, revenge or a reaction from others (4) Mostly to end or stop the pain (you couldn't go on |
| (2) Mostly to get attention, revenge or a reaction from others living with the pain or how you were feeling) |
| (3) Equally to get attention, revenge or a reaction from others (5) Completely to end or stop the pain (you couldn't go |
| on |
| and to end/stop the pain living with the pain or how you were feeling) |
| (0) Does not apply |

| SUICIDAL BEHAVIOR | Since |
|---|---|
| (Check all that apply, so long as these are separate events; must ask about all types) | Last Visit |
| Actual Attempt: | Yes No |
| A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part | ППП |
| thought of as method to kill oneself. Intent does not have to be 100%. If there is <b>any</b> intent/desire to die associated | |
| with the act, then it can be considered an actual suicide attempt. There does not have to be any injury or | Total # of |
| <i>harm</i> , just the potential for injury or harm. If person pulls trigger while gun is in mouth but gun is broken so no | Attempts |
| injury results, this is considered an attempt. | l |
| Inferring Intent: Even if an individual denies intent/wish to die, it may be inferred clinically from the behavior or | |
| circumstances. For example, a highly lethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping from window of a high floor/story). Also, if someone denies intent to die, but | Yes No |
| they thought that what they did could be lethal, intent may be inferred. | |
| Have you made a suicide attempt? | |
| Have you done anything to harm yourself? | |
| Have you done anything dangerous where you could have died? | |
| What did you do? | |
| Did you as a way to end your life? | |
| Did you want to die (even a little) when you? | |
| Were you trying to end your life when you? | |
| Or did you think it was possible you could have died from? | |
| Or did you do it purely for other reasons / without ANY intention of killing yourself (like to | |
| relieve stress, feel better, get sympathy, or get something else to happen)? (Self-Injurious | |
| Behavior without suicidal intent) | |
| If yes, describe: | |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? | |
| Interrupted Attempt: | Yes No |
| When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for | ППП |
| that, actual attempt would have occurred). | |
| Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt. Shooting: Person has gun pointed toward self, gun is taken away by | Total # of |
| someone else, or is somehow prevented from pulling trigger. Once they pull the trigger, even if the gun fails to fire, it | interrupted |
| is an attempt. Jumping: Person is poised to jump, is grabbed and taken down from ledge. Hanging: Person has | |
| noose around neck but has not yet started to hang - is stopped from doing so. | |
| Has there been a time when you started to do something to end your life but someone or | |
| something stopped you before you actually did anything? | |
| If yes, describe | |

AMX-0035 in ALS

Protocol Number: AMX3500


| Aborted Attempt: | Yes No |
|---|---|
| When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of being stopped by something else. | |
| | Total # of |
| Has there been a time when you started to do something to try to end your life but you | aborted |
| stopped yourself before you actually did anything? | |
| If yes, describe: | |
| Preparatory Acts or Behavior: | Yes No |
| Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization | |
| or thought, such as assembling a specific method (e.g., buying pills, purchasing a gun) or preparing for one's death | |
| by suicide (e.g., giving things away, writing a suicide note). | |
| Have you taken any steps towards making a suicide attempt or preparing to kill yourself | |
| (such as collecting pills, getting a gun, giving valuables away or writing a suicide note)? | |
| If yes, describe: | |
| Suicidal Behavior: | Yes No |
| Suicidal behavior was present during the assessment period? | |
| | Yes No |
| Suicide: | Yes No |
| Answer for Actual Attempts Only | Most Lethal |
| Answer for Actual Attempts Only | Most Lethal<br>Attempt |
| Answer for Actual Attempts Only | |
| Answer for Actual Attempts Only Actual Lethality/Medical Damage: | Attempt |
| | Attempt |
| Actual Lethality/Medical Damage: | Attempt<br>Date: |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second- | Attempt<br>Date: |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). | Attempt<br>Date: |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose | Attempt<br>Date: |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major | Attempt<br>Date: |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). | Attempt<br>Date: |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; | Attempt<br>Date: |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). | Attempt<br>Date: |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death | Attempt<br>Date: |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death Potential Lethality: Only Answer if Actual Lethality=0 | Attempt Date: Enter Code |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical | Attempt<br>Date: |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no | Attempt Date: Enter Code |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). | Attempt Date: Enter Code |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). 0 = Behavior not likely to result in injury | Attempt Date: Enter Code |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). | Attempt Date: Enter Code |


## 13.5 APPENDIX V: CENTER FOR NEUROLOGICAL STUDY – LABILITY SCALE

## **INSTRUCTIONS**

The purpose of this questionnaire is to help us better understand your neurologic problems. Please read each statement, and using the scale below, determine the degree to which it has applied to you **DURING THE PAST WEEK**. Circle the appropriate answer, or if you need help in marking your responses, tell the interviewer the number of the best response. Please choose only one response for each item.

| Please select the number that describes the degree to which each item has applied to you DURING THE PAST WEEK. | | | | | |
|---|---|---|---|---|---|
| | Does not<br>Apply<br>1 | Rarely<br>Applies<br>2 | Occasionally Applies 3 | Frequently Applies 4 | Applies Most of the Time 5 |
| 1. There are times when I feel fine 1 minute, and then I'll become tearful the next over something small or for no reason at all. | 0 | 0 | 0 | 0 | 0 |
| 2. Others have told me that I seem to become amused very easily or that I seem to become amused about things that aren't funny. | 0 | 0 | 0 | 0 | 0 |
| 3. I find myself crying very easily. | 0 | 0 | 0 | 0 | 0 |
| 4. I find that even when I try to control my laughter, I am often unable to do so. | 0 | 0 | 0 | 0 | 0 |
| 5. There are times when I won't be thinking of anything happy or funny at all, but then I'll suddenly be overcome by funny or happy thoughts. | 0 | 0 | 0 | 0 | 0 |
| 6. I find that even when I try to control my crying, I am often unable to do so. | 0 | 0 | 0 | 0 | 0 |
| 7. I find that I am easily overcome by laughter. | 0 | 0 | 0 | 0 | 0 |
| Evaluator's Initials: | | I. | I . | Total: | |

AMX-0035 in ALS

Protocol Number: AMX3500


### 13.6 APPENDIX VI: INSTRUCTIONS TO PATIENTS

The following instructions will be provided orally to the patient at the Baseline Visit by a healthcare staff member. Please have the Listerine® products (Pocketpaks® and Pocketmist®) available for demonstration.

- Alert the patient that the study drug has a strong bitter taste, but that there are ways to make it more palatable (see below).
- Rip open the sachet of study drug and add it to a cup or other container and add approximately 8 oz. (1 cup) of room temperature water and stir vigorously. Study drug may require significant stirring or gentle crushing to dissolve.
- The treatment should be taken within one hour of mixing into water.
- Several things may be done to reduce the bad taste and make the drug more palatable:
  - 1) Use Listerine Pocket Packs® (strips) or a Listerine PocketMist® (spray) immediately before and/or immediately after taking the drug. Use liberally to coat the mouth. This has been found to significantly mask the bitter taste.
  - 2) Take a snack or a meal after taking your treatment.
  - 3) Follow drug immediately with milk to remove taste from the mouth.
  - 4) Avoid drinking fruit juice at the same time as the drug as this may make flavor worse.
- Mixing the study drug with a liquid other than water should be avoided.








# 13.7 APPENDIX VII: AMX-0035 IN ALS OPEN LABEL EXTENSION (OLE):

## OPEN LABEL EXTENSION SCHEDULE OF ACTIVITIES

| TEN CABEL E2 | 1121(01) | | | | 7 01 1: | | 11120 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Study Drug Administration (weeks) | | | | | | Week | Week | Week | |
| ACTIVITY | Screenin<br>g/<br>Baseline<br>Visit | Wee<br>k 6 | Wee<br>k 12 | Wee<br>k 24 | Week<br>36 | Week<br>52 | Week<br>68* | Week<br>84* | 100 | 116 | 132* OR Early Discontinuati on/ Final Safety Visit |
| | Clinic | | | | | | Clinic** | | | | |
| | Day 0 <sup>8</sup> | Day<br>42<br>±10 | Day<br>84<br>±10 | Day<br>168<br>±28 | Day<br>252<br>±28 | Day<br>364<br>±28 | Day<br>476<br>±28 | Day<br>588<br>±28 | Day<br>700<br>±28 | Day<br>812<br>±28 | Day<br>924<br>±28 |
| Written Informed<br>Consent | X | | | | | | | | | | |
| Inclusion/Exclusion<br>Review | X | | | | | | | | | | |
| Vital Signs <sup>1***</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Blood Draw for<br>Safety Labs <sup>2***</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Blood Draw for<br>Serum Pregnancy<br>Test for WOCB <sup>2</sup> | X | | | | | | | | | | |
| Blood draw for<br>optional DNA<br>collection | X <sup>3</sup> | X <sup>3</sup> | X <sup>3</sup> | X <sup>3</sup> | X <sup>3</sup> | $X^3$ | X <sup>3</sup> | X <sup>3</sup> | $X^3$ | X <sup>3</sup> | X³ |
| Urine Sample for Urinalysis <sup>2***</sup> | X | X | X | X | X | X | X | X | X | X | X |
| 12-Lead ECG <sup>4***</sup> | X | X | X | X | X | X | X | X | X | X | X |
| ALSFRS-R | X | X | X | X | X | X | X | X | X | X | X |
| Slow Vital Capacity ATLIS | X<br>X | X | X | X | X | X | X | X | X | X | X<br>X |
| Columbia-Suicide<br>Severity Scale <sup>5</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Adverse Events <sup>6</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant Medications | X | Α | Λ | Λ | Α | A | A | A | A | Α | Α |
| Dispense Study<br>Drug <sup>7</sup> | X | X | X | X | X | X | X | X | X | X | |
| Key Study Events | X | X | X | X | X | X | X | X | X | X | X |
| Drug Accountability/<br>Compliance | | X | X | X | X | X | X | X | X | X | X |

Vital signs include systolic and diastolic pressure in mmHg, respiratory rate/minute, heart rate/minute, temperature and weight. Vital signs only need to be taken if they were not already recorded as part of a standard of care visit that occurred within the study visit window.

AMX-0035 in ALS

Protocol Number: AMX3500

 $Version\ 7.0$ 

<sup>&</sup>lt;sup>2</sup> Safety labs include Hematology (CBC with differential), Complete Chemistry Panel, Liver Function Tests and Urinalysis. Serum pregnancy testing will occur in women of child bearing potential (WOCBP) at the Screening Visit and as necessary during the course of the study. Blood draws and urine samples will only be taken if they were not already recorded as part of a standard of care visit that occurred within the study visit window.

- <sup>3</sup> Optional one-time blood draw for DNA analysis can be completed during the OLE, if not completed during main study.
- 4 12-Lead ECG only needs to be completed if it was not already recorded as part of a standard of care visit that occurred within the study visit window.
- <sup>5</sup> C-SSRS Since Last Visit version to be completed at all visits.
- <sup>6</sup> Adverse events that are ongoing from the main study should be recorded and followed during the OLE. Any new adverse events that occur AFTER start of OLE treatment will be recorded.
- <sup>7</sup> First dose of study drug will be administered in clinic after ALL Screening/Baseline Visit procedures are completed.
- 8 Day 0 Visit of the open label extension sub-study may be the same as Week 24 Visit of the main study so that exams and tests do not need to be duplicated if the Day 0 visit occurs within 7 days of the Week 24 visit. If the subject enrolls day 8-28 then all assessments for the Day 0 visit should be completed. Subjects must enroll in the OLE within 28 days of the Week 24 visit of the main study.
- \* If subject is unable to complete all procedures, minimal procedures should be completed in the following suggested order: ALSFRS-R, AE Review, Safety labs, ECG, Concomitant Medication.
- \*\* Study visits may occur remotely. If possible, remote visits should be conducted using a HIPAA-compliant video conferencing platform. If video conferencing is not available or not feasible, remote visits may be conducted by phone. If the visit is not conducted in person, the following procedures should be completed in the following suggested order: ALSFRS-R, AE Review, Key Study Event, Concomitant Medications, Columbia-Suicide Severity Scale, and Dispense Study Drug. Drug product will be dispensed to subjects only after the SI has reviewed the necessary safety procedures for the subject to take the study drug.
- \*\*\* In order for subject to remain on study drug, these procedures must be performed every six (6) months to monitory safety. These procedures can be done during a clinic visit at the study site or done remotely using a local health facility or home nurse service. Interim safety procedures can be done at each study visit, at the discretion of the SI.

AMX-0035 in ALS Protocol Number: AMX3500 Version 7.0 Version date 30Mar2020

## **OPEN LABEL EXTENSION PLAN**

## **Study Indication**

Amyotrophic Lateral Sclerosis (ALS)

# **Phase of Development**

II

## **Rationale for the Study**

The objective of this study is to determine the long-term safety of AMX0035 in subjects with Amyotrophic Lateral Sclerosis (ALS). ALS is a progressive neurodegenerative disease for which there is no cure. There are only two medicines approved specifically for treating ALS, Rilutek (riluzole) and Radicava (edaravone). ALS also exacts a significant economic burden.

AMX0035 has demonstrated efficacy in models of neurodegeneration, classical activation of neuroinflammation, and bioenergetics deficits. The individual components of AMX0035, PB and TUDCA have demonstrated efficacy in in vivo models of ALS, Parkinson's, Alzheimer's, ischemia, and many others. Each individual component has also been tested in small clinical trials of ALS subjects and was found to be safe and well-tolerated, and hit primary endpoints of efficacy.

## **Study Design and Plan**

This is a multicenter, open label extension, up to 132-week study evaluating the long-term safety of AMX0035. Up to one hundred thirty-two (132) subjects will be given oral (or feeding tube) twice daily sachet of active therapy. Treatment duration will be up to one thirty-two (132) weeks starting at the Screening/Baseline visit. Clinic visits will occur at Screening/Baseline, Week 6 (day 42), Week 12 (day 84), Week 24 (day 168), Week 36 (day 252), and Week 52 (Day 364), Week 68 (Day 476), Week 84 (Day 588), Week 100 (Day 700), Week 116 (Day 812), Week 132 (Day 924). Study visits may occur remotely, as needed. If possible, remote visits should be conducted using a HIPAA-compliant video conferencing platform. If video conferencing is not available or not feasible, remote visits may be conducted by phone. If the visit is not conducted in person, the following procedures should be completed in the following suggested order: ALSFRS-R, AE Review, Key Study Event, Concomitant Medications, Columbia-Suicide Severity Scale.

All visit windows are consecutive calendar days and are calculated from the day the subject starts study treatment (Day 0, the day of the Screening/Baseline Visit). The screening/Baseline visit must occur within 28 days of the Week 24 visit of the main study. If the Screening/Baseline visit occurs on the day of the Week 24 visit or within 7 days of that visit then it is not necessary to complete the assessments, labs and outcomes. If the Screening/Baseline visit occurs Day 8 – Day 28 then all assessments, labs and outcomes need to be completed. Visit windows will be +/- 10 days for the Week 6 and Week 12 visits and +/- 28 days for the Week 24, Week 36, Week 52, Week 68, Week 84, Week 100, Week 116 and Week 132 visits. Any change from this visit window will be considered an out of window visit deviation.


## **Study Objectives**

The primary objective of the study is to assess long-term safety of oral (or feeding tube) administration of AMX0035 via sachet (3g PB and 1g TUDCA) twice daily for compassionate use.

The primary outcome measure is:

1. To confirm the long-term safety of AMX0035 in subjects with ALS over a 132-week period

Secondary outcome measures will include:

- 1. The rate of key study events including tracheostomy, hospitalization, and death
- 2. Rate of progression on the ALSFRS-R scale
- 3. ATLIS rate of progression
- 4. Rate of progression of slow vital capacity

## **Study Locations**

Up to 25 Northeast ALS Consortium (NEALS) centers in the United States that participated in the randomized, double-blind trial will participate in this study.

## **Number of Planned Subjects**

Up to 132 subjects that participated in the randomized, double-blind trial will be able to enroll in this study.

## **Study Population**

This study will be conducted in subjects who have sporadic or familial ALS diagnosed as definite as defined by revised El Escorial criteria (Appendix 1). Subjects must provide written informed consent prior to screening. At screening/baseline subjects must have completed participation in the randomized, double-blind trial.

### **Study Enrollment**

Inclusion Criteria:

- 1. Completion of all visits in the randomized, double blind AMX0035 study. Subjects that receive tracheostomy or PAV during the course of the main study will still be followed as ITT until the week 24 visit before enrollment in the OLE.
- 2. Must enroll in the OLE within 28 days of the Week 24 visit of the main study.
- 3. Signed informed consent to enter the open label extension phase.

### Exclusion Criteria:

- 1. Discontinued study drug prematurely in the double-blind phase of the study for reasons other than tracheostomy or PAV.
- 2. Exposure to or anticipated requirement for any disallowed medication listed below.
- 3. Any ongoing adverse events that in the opinion of the Site Investigator are clear contraindications to the study drug.
- 4. Unstable cardiac or other life-threatening disease emergent during the randomized, double blind study

AMX-0035 in ALS Protocol Number: AMX3500


5. Any major medical condition that in the opinion of the Site Investigator would interfere with the study and place the subject at increased risk.

Subjects who receive tracheostomy or PAV while in the randomized, double-blind trial can elect to enroll in the OLE so long as they complete all visits in the main study.

Disallowed medications for all subjects include:

- HDAC Inhibitors including:
  - o Valproate
  - Vorinostat (Zolinza)
  - o Romidepsin
  - o Chidamide
  - o Panobinostat
  - o Lithium
  - o Butyrate
  - o Suramin
- Probenecid
- Bile Acid Sequestrants including:
  - o Cholestyramine and Cholestyramine Light
  - o Questran and Questran Light
  - Welchol
  - o Colestid and Colestid Flavored
  - o Prevalite

# Note on Antacids Within Two Hours of Study Drug Administration

Antacids containing Aluminum hydroxide or smectite (aluminum oxide) may not be taken within two hours of administration of the study drug as they inhibit absorption of TUDCA.

#### These include:

- o Alamag
- o Alumina and Magnesia
- o Antacid, Antacid M and Antacid Suspension
- o Gen-Alox
- Kudrox
- o M.A.H.
- o Maalox HRF and Maalox TC
- Magnalox
- o Madroxal
- o Mylanta and Mylanta Ultimate
- o Ri-Mox

AMX-0035 in ALS

Protocol Number: AMX3500

 $Version\ 7.0$ 

#### $\circ$ Rulox

Please refer to section 6.7 and 6.7.1 of the main protocol for all medication information.

# **Study Drug and Treatment Administration**

There will be a new formulation for the open label extension that has been optimized for better taste.

A powder filled sachet will be used as the AMX0035 drug product. The drug product will be filled under cGMP conditions in an aluminum foil lined sachet.

The sachet containing active ingredients will include:

- o Active Ingredients:
  - 1g TUDCA
  - 3g PB (Phenylbutyrate)
- Excipients
  - Dextrates
  - Sorbitol
  - Sucralose
  - Syloid 63FP (colloidal silica)
  - Kleptose Linecaps (maltodextrin)
  - Firmenich Flavor Masking Flavorant
  - Firmenich Mixed Berry Flavorant
  - Sodium Phosphate Dibasic
  - Sodium Stearyl Fumarate

Changes from the batch used in the randomized, double blind study include a different level of sucralose, the mixed berry flavor being provided by a new company and the addition of a flavor masking agent.

Please see section 6 of the main protocol for more information on the description, packaging, storage, dosage, administration, concomitant therapies and prohibited medications of the study drug.

Study drug will be provided in clinic on the day of the screening/baseline visit and re-supplied at each subsequent visit.

Subjects should bring in unused sachets so that the site may check compliance. Any unused sachets should be re-dispensed to the subject during the visit. Please refer to the site MOP for a detailed description of study drug dispensing.

Subjects will take 2 sachets daily, 1 sachet in the morning and 1 sachet in the afternoon, throughout the study.


In order for subjects to remain on study drug, the following safety procedures must continue to be performed every six (6) months to monitor safety. Interim safety procedures can be done at each study visit, at the discretion of the SI. These procedures can be done during the clinic visit or remotely using a local health facility or home nurse service:

- 1. Vital signs including blood pressure, body weight, and temperature
- 2. 12-lead ECG (Electrocardiogram)
- 3. Laboratory assessments including Hematology (CBC with differential), Complete Chemistry Panel, Liver Function Tests
- 4. Urinalysis

## **Duration of Treatment and Follow-up**

Subjects will remain on treatment until the Week 132 or early discontinuation visit.

## **Study Schedule**

No study procedures should be performed prior to the signing of the informed consent form (ICF). All subjects will sign an ICF prior to undergoing any study tests or procedures. To the extent possible, the Schedule of Activities for each study visit should be performed. It is recommended that the ALSFRS-R and ATLIS are completed first at each study visit and Blood Samples are drawn at the end of the study visit. If subject is unable to complete all procedures during the in-person clinic study visits, minimal procedures should be completed in the following suggested order: ALSFRS-R, AE Review, Safety Labs, ECG, and Concomitant Medications.

Study visits may occur remotely as needed. If possible, remote visits should be conducted using a HIPAA-compliant video conferencing platform. If video conferencing is not available or not feasible, remote visits may be conducted by phone. If the visit is not conducted in person, the following procedures should be completed in the suggested order: ALSFRS-R, AE Review, Key Study Event, Concomitant Medications, Columbia-Suicide Severity Scale.

Visit windows are consecutive calendar days and the target visit dates are calculated from the Screening/Baseline Visit.

Subjects who withdraw consent or early terminate from the study (i.e., discontinue study drug) will be asked to come in for a Final Safety Visit.

# Screening/Baseline Clinic Visit:

Day 0 Visit of the open label extension sub-study may be the same as Week 24 Visit of the main study - so that exams and tests do not need to be duplicated if they were previously completed.

The following procedures will be performed:

- Obtain written informed consent from subject
- o Assess inclusion and exclusion criteria
- o Review and document concomitant medications and therapies


- Administer C-SSRS (Baseline Version)
- o Administer ALSFRS-R questionnaire
- o Measure isometric strength using ATLIS machine
- o Assess and document adverse events (AEs) that occur after subject signs informed consent form (ICF)
- o Measure vital signs (blood pressure, heart and breathing rates, temperature, and weight)
- o Perform 12-lead ECG (Electrocardiogram)
- o [After other tests] Collect blood samples for clinical laboratory assessments including Hematology (CBC with differential), Complete Chemistry Panel, Liver Function Tests, serum pregnancy test (for women of child-bearing potential [WOCBP]), optional DNA analysis if not completed during main study
- o Collect urine sample for urinalysis
- O Dispense 2 kits of study drug (12 weeks + 2 weeks extra)
- o Capture key study events
- o Schedule the Week 6 Visit

# Week 6, Week 12, Week 24, Week 36, Week 52, Week 68, Week 84, Week 100, Week 116, Week 132 or Early Discontinuation/Final Safety Clinic Visit:

The Week 6 and Week 12 visits will take place +/- 10 days and the Week 24, Week 36, Week 52, Week 68, Week 84, Week 100, Week 116 and Week 132 visits will take place +/- 28 days from the time specified in the schedule of activities (table as beginning of this section).

The following procedures will be performed:

- o Review and assess Adverse Events
- Measure vital signs
- o Administer the C-SSRS questionnaire (Since Last Visit)
- o Administer ALSFRS-R questionnaire
- o Measure isometric strength using ATLIS machine
- o Perform 12-lead ECG (Electrocardiogram)
- Collect blood samples for clinical laboratory assessments including Hematology (CBC with differential), Complete Chemistry Panel, Liver Function Tests, optional DNA analysis if not completed during main study
- o Collect urine sample for urinalysis
- o Perform study drug accountability
- o Dispense study drug (Except at Week 132/Early Discontinuation)
- o Capture key study events
- o Schedule next study visit (Except Week 132/Early Discontinuation)

Please note – safety labs, urine collection for urinalysis, pregnancy test, and 12-lead ECG do not need to be repeated if they were completed as part of clinical or SOC visit within the approved study visit window.


# **Laboratory Testing:**

The following laboratory tests will be performed for safety:

- Hematology with differential panel: complete blood count with differential (hematocrit, hemoglobin, platelet count, RBC indices, Total RBC, Total WBC, and WBC & differential)
- Blood chemistry panel/Liver function tests (LFTs): alanine aminotransferase (ALT (SGPT)), aspartate aminotransferase (AST (SGOT)), albumin, alkaline phosphatase, bicarbonate, blood urea nitrogen, calcium, chloride, creatinine, glucose, potassium, sodium, total bilirubin and total protein
- o Urinalysis:, bilirubin, blood, clarity, color, glucose, ketones, nitrate, pH, protein, specific gravity, urobilinogen and WBC screen
- Serum human chorionic gonadotrophin (hCG) for women of childbearing potential (WOCBP) (collected only at Screening Visit, and as necessary throughout course of study)

Please note: for the OLE portion of the study, local laboratories will be used.

In order for subjects to remain on study drug, laboratory testing must continue to be performed every six (6) months to monitor safety. Interim laboratory testing can be done at each study visit, at the discretion of the SI. This laboratory testing can be done remotely using a local health facility or home nurse service, if clinic visit is not feasible.

## **Safety and Adverse Events**

For the purposes of this study, an adverse event (AE) will be defined as any unfavorable and unintended sign, symptom, or disease that the Site Investigator deems to be definitely, probably, possibly, unlikely or not related to the conduct of the study procedures or study drug.

Please refer to section 9 of the main protocol for more information on adverse events.

## **Data Safety and Monitoring and Statistical Analysis Plan**

Please refer to section 7.16 and 7.17 regarding protocol deviations, missed visits and deaths. Please refer to section 9 of this protocol regarding safety management. The safety management plan contains additional details regarding safety management. Please refer to section 11 regarding data capture. A separate statistical analysis plan will be prepared for this study.

Statistical analysis will mainly entail analysis of types and frequencies of adverse events. Measures of SVC, ATLIS, ALSFRS-R and study events in the open label extension study will be compared to the double-blind

AMX-0035 in ALS Protocol Number: AMX3500 Version 7.0 Version date 30Mar2020 section of this study and to historical data. A detailed description of the statistical plan is contained in the section titled, "Open Label Extension Statistical Analysis Plan."

While the blinded study is ongoing, the DSMB will review safety events in this study during its regular meeting, as detailed in the DSMB charter. When the main study is concluded (last patient out), the independent Medical Monitor will review ongoing safety for the remainder of the extension.

AMX-0035 in ALS Protocol Number: AMX3500 Version 7.0 Version date 30Mar2020